| Stay Connected: Testing an | Intervention to Comba | at COVID-19 Related | Social Isolation | Among Seattle- |
|---|---|---|---|---|
| | area Olo | der Adults | | |

NCT04966910

3/11/2021



The Human Subjects Division (HSD) strives to ensure that people with disabilities have access to all services and content. If you experience any accessibility-related issues with this form or any aspect of the application process, email <a href="https://hsd.nico.new.edu">hsdinfo@uw.edu</a> for assistance.

#### **INSTRUCTIONS**

- This form is only for studies that will be reviewed by the UW IRB. Before completing this form, check HSD's website to confirm that this should not be reviewed by an external (non-UW) IRB.
- <u>If you are requesting a determination</u> about whether the planned activity is human subjects research or qualifies for exempt status, you may skip all questions except those marked with a . For example 1.1 must be answered.
- Answer all questions. If a question is not applicable to the research or if you believe you have already answered a question elsewhere in the application, state "NA" (and if applicable, refer to the question where you provided the information). If you do not answer a question, the IRB does not know whether the question was overlooked or whether it is not applicable. This may result in unnecessary "back and forth" for clarification. Use non-technical language as much as possible.
- To check a box, place an "X" in the box. To fill in a text box, make sure your cursor is within the gray text box bar before typing or pasting text.
- For collaborative or multi-site research, describe only the UW activities unless you are requesting that the UW IRB provide the review and oversight for non-UW collaborators or co-investigators as well.
- You may reference other documents (such as a grant application) if they provide the requested information in non-technical language. Be sure to provide the document name, page(s), and specific sections, and upload it to *Zipline*. Also, describe any changes that may have occurred since the document was written (for example, changes that you've made during or after the grant review process). In some cases, you may need to provide additional details in the answer space as well as referencing a document.

| INDEX | | |
|---|---|---|
| 1 Overview | 6 Children (Minors) and Parental Permission | 10 Risk / Benefit Assessment |
| 2 Participants | 7 Assent of Children (Minors) | 11 Economic Burden to Participants |
| 3 Non-UW Research Setting | 8 Consent of Adults | 12 Resources |
| 4 Recruiting and Screening Participants | 9 Privacy and Confidentiality | 13 Other Approvals, Permissions, and<br>Regulatory Issues |
| 5 Procedures | | |

APPLICATION IRB Protocol

# **1 OVERVIEW**

**Study Title:** 

Stay Connected: Co-design and testing an intervention to combat COVID-19 related social isolation among Seattle-area seniors

(1.1) Home institution. Identify the institution through which the lead researcher listed on the IRB application will conduct the research. Provide any helpful explanatory information.

In general, the home institution is the institution (1) that provides the researcher's paycheck and that considers him/her to be a paid employee, or (2) at which the researcher is a matriculated student. Scholars, faculty, fellows, and students who are visiting the UW and who are the lead researcher: identify your home institution and describe the purpose and duration of your UW visit, as well as the UW department/center with which you are affiliated while at the UW.

Note that many UW clinical faculty members are paid employees of non-UW institutions.

The UW IRB provides IRB review and oversight for only those researchers who meet the criteria described in the **SOP: Use of the UW IRB**.

University of Washington

(1.2)Consultation history. Has there been any consultation with someone at HSD about this study?

It is not necessary to obtain advance consultation. However, if advance consultation was obtained, answering this question will help ensure that the IRB is aware of and considers the advice and guidance provided in that consultation.



→ If yes, briefly describe the consultation: approximate date, with whom, and method (e.g., by email, phone call, in-person meeting).

Phone Call with Bailey Bodell

(1.3) Similar and/or related studies. Are there any related IRB applications that provide context for the proposed activities?

Examples of studies for which there is likely to be a related IRB application: Using samples or data collected by another study; recruiting subjects from a registry established by a colleague's research activity; conducting Phase 2 of a multi-part project, or conducting a continuation of another study; serving as the data coordinating center for a multi-site study that includes a UW site.

Providing this information (if relevant) may significantly improve the efficiency and consistency of the IRB's review.



→ If yes, briefly describe the other studies or applications and how they relate to the proposed activities. If the other applications were reviewed by the UW IRB, please also provide: the UW IRB number, the study title, and the lead researcher's name.

STUDY00010021 was the first phase of this project, a survey of Seattle-area senior housing residents and middle-school students, about the impact of COVID-19 related social isolation. This protocol represents the next steps in that project with older adults.

**1.4** Externally-imposed urgency or time deadlines. Are there any externally-imposed deadlines or urgency that affect the proposed activity?

HSD recognizes that everyone would like their IRB applications to be reviewed as quickly as possible. To ensure fairness, it is HSD policy to review applications in the order in which they are received. However, HSD will assign a higher priority to research with externally-imposed urgency that is beyond the control of the researcher. Researchers are encouraged to communicate as soon as possible with their HSD staff contact person when there is an urgent situation (in other words, before submitting the IRB application). Examples: a researcher plans to test an experimental vaccine that has just been developed for a newly emerging epidemic; a researcher has an unexpected opportunity to collect data from students when the end of the school year is only four weeks away.

HSD may ask for documentation of the externally-imposed urgency. A higher priority should not be requested to compensate for a researcher's failure to prepare an IRB application in a timely manner. Note that IRB review requires a certain minimum amount of time; without sufficient time, the IRB may not be able to review and approve an application by a deadline.



→ If yes, briefly describe the urgency or deadline as well as the reason for it.

We have received a NIMH supplement to Dr. Arean's ALACRITY Center to support this work. IRB approval is required prior to receipt of the funds.

(1.5) Objectives Using lay language, describe the purpose, specific aims, or objectives that will be met by this specific project. If hypotheses are being tested, describe them. You will be asked to describe the specific procedures in a later section.

If this application involves the use of a HUD "humanitarian" device: describe whether the use is for "on-label" clinical patient care, "off-label" clinical patient care, and/or research (collecting safety and/or effectiveness data).

COVID-19 pandemic social distancing practices have the following unintended consequences for have older adults living in senior housing facilities and independent living communities: social isolation, loneliness, depression, and anxiety. Staff at these facilities likewise struggle with managing social distance practices and the well-being of their residents. We propose to co-design a lay-worker delivered intervention with older adults and housing staff members or administrators. We will demonstrate a number of potential programs and activities to reduce social isolation and enhance cognitive stimulation and emotional well-being such as Patient Activation, anxiety management, virtual social support groups, activities to connect public school students (another social isolation risk group) and emerging on-line tools such as remote concerts and on-line learning. Reactions and suggestions will be collected, and participants will help co-design the beta version the "Stay Connected" intervention package that we will test in a pilot RCT. Intended outcomes will be social connection, self-efficacy in coping with social isolation, symptoms of depression and health-related anxiety.

(1.6) Study design. Provide a one-sentence description of the general study design and/or type of methodology.

Your answer will help HSD in assigning applications to reviewers and in managing workload. Examples: a longitudinal observational study; a double-blind, placebo-controlled randomized study; ethnographic interviews; web scraping from a convenience sample of blogs; medical record review; coordinating center for a multi-site study.

Design/Build Phase: Co-design a lay-worker delivered intervention with older adults and housing staff members or administrators

Test Phase: Pilot, proof of concept randomized control trial of the "Stay Connected" intervention. We will submit a modification for Test Phase procedures after completion of the Design/Build phase.

**1.7** Intent. Check all the descriptors that apply to your activity. You must place an "X" in at least one box.

This question is essential for ensuring that your application is correctly reviewed. Please read each option carefully.

| Descriptor |
|---|
| Class project or other activity whose purpose is to provide an educational experience for the researcher (for example, to learn about the process or methods of doing research). |
| 2. Part of an institution, organization, or program's own internal operational monitoring. |
| 3. Improve the quality of service provided by a specific institution, organization, or program. |
| <ul> <li>4. Designed to expand the knowledge base of a scientific discipline or other scholarly field of study, and produce results that: <ul> <li>Are expected to be applicable to a larger population beyond the site of data collection or the specific subjects studied, or</li> <li>Are intended to be used to develop, test, or support theories, principles, and statements of relationships, or to inform policy beyond the study.</li> </ul> </li> </ul> |
| 5. Focus directly on the specific individuals about whom the information or biospecimens are collected through oral history, journalism, biography, or historical scholarship activities, to provide an accurate and evidence-based portrayal of the individuals. |
| 6. A quality improvement or program improvement activity conducted to improve the implementation (delivery or quality) of an accepted practice, or to collect data about the implementation of the practice for clinical, practical, or administrative purposes. This does not include the evaluation of the efficacy of different accepted practices, or a comparison of their efficacy. |
| 7. Public health surveillance activities conducted, requested, or authorized by a public health authority for the sole purpose of identifying or investigating potential public health signals or timely awareness and priority setting during a situation that threatens public health. |
| 8. Preliminary, exploratory, or research development activities (such as pilot and feasibility studies, or reliability/validation testing of a questionnaire) |
| 9. Expanded access use of a drug or device not yet approved for this purpose |
| 10. Use of a Humanitarian Use Device |
| 11. Other. Explain: |

- **1.8 Background, experience, and preliminary work**. Answer this question <u>only</u> if the proposed activity has one or more of the following characteristics. The purpose of this question is to provide the IRB with information that is relevant to its risk/benefit analysis.
  - Involves more than minimal risk (physical or non-physical)
  - Is a clinical trial, or
  - Involves having the subjects use a drug, biological, botanical, nutritional supplement, or medical device.

"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

**a.** <u>Background</u>. Provide the rationale and the scientific or scholarly background for the proposed activity, based on existing literature (or clinical knowledge). Describe the gaps in current knowledge that the project is intended to address.

This should be a plain language description. Do not provide scholarly citations. Limit your answer to less than one page, or refer to an attached document with background information that is no more than three pages long.

COVID-19 pandemic social distancing practices have the following unintended consequences for have older adults living in senior housing facilities and independent living communities: social isolation, loneliness, depression, and anxiety. Staff at these facilities likewise struggle with managing social distance practices and the well-being of their residents. We intend to survey older adults and staff members about the impact of social isolation on mental health and well-being. This project intends to address the lack of understanding about the impact of COVID-19 related social isolation on these populations, and to learn directly from those impacted about potential strategies to combat the effects on mental health and well-being.

**b.** Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you, your team, or your collaborators/co-investigators have that supports the feasibility and/or safety of this study.

It is not necessary to summarize all discussion that has led to the development of the study protocol. The IRB is interested only in short summaries about experiences or preliminary work that suggest the study is feasible and that risks are reasonable relative to the benefits. Examples: Your team has already conducted a Phase 1 study of an experimental drug which supports the Phase 2 study being proposed in this application; your team has already done a small pilot study showing that the reading skills intervention described in this application is feasible in an after-school program with classroom aides; your team has experience with the type of surgery that is required to implant the study device; the study coordinator is experienced in working with subjects who have significant cognitive impairment.

We have completed a survey of Seattle-area senior housing residents and completed interviews with staff and administrators at Seattle-area senior housing facilities to learn about the impact of COVID-19 related social isolation which showed residents experiencing loneliness and at-risk of mental health concerns, including depression and anxiety. Additionally, our survey found that COVID-19 related social distancing has resulted in significant impacts on social engagement and activity levels thus supporting the need for an intervention to address depression, anxiety, and social isolation in senior living communities.

This project is a partnership between the UW CREATIV Lab and UW ALACRITY Center. The CREATIV Lab brings extensive experience working with this target population. The ALACRITY Center brings extensive experience in user-centered design and implementation of interventions in diverse settings.

**1.9 Supplements**. Check all boxes that apply, to identify relevant Supplements that should be completed and uploaded to *Zipline*.

This section is here instead of at the end of the form to reduce the risk of duplicating information in this IRB Protocol form that you will need to provide in these Supplements.

| Check all<br>That Apply | Type of Research | Supplement Name |
|---|---|---|
| | <b>Department of Defense</b> The research involves Department of Defense funding, facilities, data, or personnel. | SUPPLEMENT Department of Defense |
| | <b>Department of Energy</b> The research involves Department of Energy funding, facilities, data, or personnel. | SUPPLEMENT Department of Energy |
| | <b>Drug, biologic, botanical, supplement</b> Procedures involve the use of <u>any</u> drug, biologic, botanical or supplement, even if the item is not the focus of the proposed research | SUPPLEMENT Drugs |
| | Emergency exception to informed consent Research that requires this special consent waiver for research involving more than minimal risk | SUPPLEMENT Exception<br>from Informed Consent<br>for Emergency Research<br>(EFIC) |
| | Genomic data sharing Genomic data are being collected and will be deposited in an external database (such as the NIH dbGaP database) for sharing with other researchers, and the UW is being asked to provide the required certification or to ensure that the consent forms can be certified | SUPPLEMENT Genomic Data Sharing |
| | Medical device Procedures involve the use of <u>any</u> medical device, even if the device is not the focus of the proposed research, except when the device is FDA-approved and is being used through a clinical facility in the manner for which it is approved | SUPPLEMENT Devices |
| | Multi-site or collaborative study The UW IRB is being asked to review on behalf of one or more non-UW institutions in a multi-site or collaborative study. | SUPPLEMENT: Multi-site<br>or Collaborative Research |
| х | Non-UW Individual Investigators The UW IRB is being asked to review on behalf of one or more non-UW individuals who are not affiliated with another organization for the purpose of the research. | SUPPLEMENT: Non-UW<br>Individual Investigators |
| | None of the above | |

(d) no participants over the age of 85 years will be enrolled. See this webpage for details, including what "screening" means.

# X Confirmed

# **2 PARTICIPANTS**

**2.1** Participants. Describe the general characteristics of the subject populations or groups, including age range, gender, health status, and any other relevant characteristics.

## Design/Build Phase

In the design/build phase, we will work with senior living residents and staff.

- (1) Older Adults: We will recruit up to 15 older adults living in senior living communities in the Seattle area. Similar to above, while we expect these these individuals to be over the age of 65, we will not limit our sample by age. The health status of these individuals will vary from no health concerns to multiple chronic health conditions. The unifying characteristic of this group is their status as a resident of a senior living community. These may be individuals that participated in the survey phase of the study.
- (2) Senior Living Community Staff: We will recruit up to 3 staff members from senior living communities in the Seattle area. The age, gender and health status of these individuals will vary and do not impact their participation in the study. These may be individuals that participated in the survey phase of the study.

#### **Test Phase**

In the test phase, we will work with senior living residents and staff.

- (1) Older Adults: We will recruit up to 120 older adults, aged 60+ from senior living communities or senior centers in the Seattle area. These participants will meet the same general characteristics as older adult participants in the Design/Build phase.
- (2) Senior Living Community or Senior Center Staff: We will recruit up to 12 staff from senior housing communities and/or senior centers in the Seattle area. As with previous phases, the age, gender, and health status of these individuals will vary and do not impact their participants in the study. These may be individuals that participated in previous phases of the study. These individuals will be study participants and they will also deliver the intervention designed in the previous phase of the study if the senior living community or senior center at which they work is randomized to Stay Connected.

# (2.2) Inclusion and exclusion criteria.

**a. Inclusion criteria.** Describe the specific criteria that will be used to decide who will be included in the research from among interested or potential subjects. Define any technical terms in lay language.

#### Design/Build Phase

We will have 2 different participant groups for this phase: (1) senior living community staff and (2) older adults.

- (1) Senior Living Community Staff: English-speaking staff members in administration, social work, and/or activities departments at Seattle-area senior living communities; Physical ability to complete interviews over the phone or using video-based technology (ex. Zoom); Cognitive ability to consent and complete interviews
- (2) Older Adults: English-speaking residents of Seattle-area senior living communities; Physical and cognitive ability to complete interviews by phone or using video-chat technology (ex. Zoom); Ability to provide consent

#### Test Phase

In the test phase, we will have two different participant groups: (1) Senior Living Community Staff and (2) Older Adults:

- (1) Senior Living Community or Senior Center Staff: English-speaking staff members in administration, social work, and/or activities departments at Seattle-area senior living communities; Physical ability to complete training in intervention and complete questionnaires by phone, computer, or video-chat technology
- (2) Older Adults: English-speaking residents of Seattle-area senior living communities or members of senior centers; 60 years old and older; Physical and cognitive ability to complete interviews by phone or using video-chat technology (ex. Zoom); Ability to provide consent; Scores of 5 or higher on PHQ-9 OR Score of 5 or higher on GAD-7 OR 6 or higher on UCLA Loneliness Scale; No active suicidal ideation
- **b. Exclusion criteria.** Describe the specific criteria that will be used to decide who will be excluded from the research from subjects who meet the inclusion criteria listed above. Define any technical terms in lay language.

#### Design/Build Phase

We will have 2 different participant groups for this phase: (1) senior living community staff and (2) older adults.

- (1) Senior Living Community Staff: Non-English speaking; Unable to physically or cognitively consent and/or participate in study procedures via phone, computer, and/or video call (e.g. Zoom)
- (2) Older Adults: Non-English speaking; Under the age of 60; Unable to physically or cognitively consent and/or participate in study procedures via phone, computer, and/or video call (e.g. Zoom)

#### Test Phase

We will have 2 different participant groups for this phase: (1) senior living community staff and (2) older adults.

- (1) Senior Living Community or Senior Center Staff: Non-English speaking; Unable to physically or cognitively consent and/or participate in study procedures via phone, computer, and/or video call (e.g. Zoom)
- (2) Older Adults: Non-English speaking; Under the age of 60; Unable to physically or cognitively consent and/or participate in study procedures via phone, computer, and/or video call (e.g. Zoom); Active suicidal ideation; Scores below inclusion cut offs on PHQ-9, GAD-7, and UCLA Loneliness Scale
- **2.3 Prisoners**. IRB approval is required in order to include prisoners in research, even when prisoners are not an intended target population.
  - a. Will the proposed research recruit or obtain data from individuals that are known to be prisoners?

For records reviews: if the records do not indicate prisoner status and prisoners are not a target population, select "No". See the <u>WORKSHEET Prisoners</u> for the definition of "prisoner".

| Х | No | $\rightarrow$ If no, skip the rest of part a. and continue to 2.3.b |
|---|---|---|
| | Yes | → If yes, answer the following questions (i – iv). |

i. Describe the type of prisoners, and which prisons/jails:

| | earnings in prison will be so great | care, quality of food, amenities, and/or opportunity for that it will make it difficult for prisoners to adequately vill the chances of this be reduced? |
|---|---|---|
| | procedures will be fair to all eligib | ke sure that (a) recruitment and subject selection<br>le prisoners and (b) prison authorities or other prisoners<br>ent or require particular prisoners from participating. |
| | Washington State: check the box (a) not encourage or facilitate the influence parole decisions, and (b) | ers in federal facilities or in state/local facilities outside of below to provide assurance that study team members will use of a prisoner's participation in the research to clearly inform each prisoner in advance (for example, in a nather than the research will have no effect on his or her parole. |
| <b>b.</b> Is the resear | | ne prisoners while participating in the study? |
| point during to | he study. → If yes, if a subject becomes a prison | related to the subject be continued while the subject is a |
| | Yes → If yes, describe the p prisoner subjects | rocedures and/or data collection that will continue with |
| boxes for any of | · | e use of the subject populations listed here. Check the efully included. (In other words, being a part of the |
| The WORKSHEETS | describe the criteria for approval but do | not need to be completed and should not be submitted. |
| | Population | Worksheet |
| Fetuses in u | itero | WORKSHEET Pregnant Women |
| Neonates o | f uncertain viability | WORKSHEET Neonates |
| Non-viable | neonates | WORKSHEET Neonates |
| Pregnant w | omen | WORKSHEET Pregnant Women |

ii. One concern about prisoner research is whether the effect of participation on prisoners'

Version 2.50

| defined in international or national legislation as having a set of specific rights based on their ticular territory and their cultural or historical distinctiveness from other populations that are often school or health clinic; recruiting during a tribal community gathering, name the tribe, tribal-focused organization, or similar community-based organization. RB expects that tribal/indigenous approval will be obtained before beginning the research may or may not involve approval from a tribal IRB. The study team and any corators/investigators are also responsible for identifying any tribal laws that may affect arch. |
|---|
| , name the tribe, tribal-focused organization, or similar community-based organization. RB expects that tribal/indigenous approval will be obtained before beginning the researce may or may not involve approval from a tribal IRB. The study team and any corators/investigators are also responsible for identifying any tribal laws that may affect |
| RB expects that tribal/indigenous approval will be obtained before beginning the researd may or may not involve approval from a tribal IRB. The study team and any corators/investigators are also responsible for identifying any tribal laws that may affect |
| Will the research collect private identifiable information about other individuals from the most of |
| any direct or indirect identifier that, alone or in combination, would allow you or another member readily identify the person. For example, suppose that the research is about immigration history. I estions about their grandparents but are not asked for names or other information that would allow the grandparents, then private identifiable information is not being collected about the grandpare are not subjects. |
| es, these individuals are considered human subjects in the study. Describe them and wha |

**2.7 Number of subjects.** Is it possible to predict or describe the maximum number of subjects (or subject units) needed to complete the study, for each subject group?

<u>Subject units</u> mean units within a group. For most research studies, a group will consist of individuals. However, the unit of interest in some research is not the individual. Examples:

- Dyads such as caregiver-and-Alzheimer's patient, or parent and child
- Families
- Other units, such as student-parent-teacher

<u>Subject group</u> means categories of subjects that are meaningful for the specific study. Some research has only one subject group – for example, all UW students taking Introductory Psychology. Some common ways in which subjects are grouped include:

- By intervention for example, an intervention group and a control group.
- By subject population or setting for example, urban versus rural families
- By age for example, children who are 6, 10, or 14 years old.

The IRB reviews the number of subjects in the context of risks and benefits. Unless otherwise specified, if the IRB determines that the research involves no more than minimal risk: there are no restrictions on the total number of subjects that may be enrolled. If the research involves more than minimal risk: The number of enrolled subjects must be limited to the number described in this application. If it is necessary later to increase the number of subjects, submit a Modification. Exceeding the IRB-approved number (over-enrollment) will be considered non-compliance.

No

→ If no, provide the rationale in the box below. Also, provide any other available information about the scope/size of the research. You do not need to complete the table.

Example: It may not be possible to predict the number of subjects who will complete an online survey advertised through Craigslist, but you can state that the survey will be posted for two weeks and the number who respond is the number who will be in the study.

Yes → If yes, for each subject group, use the table below to provide the estimate of the maximum desired number of individuals (or other subject unit, such as families) who will complete the research.

| Group name/description | Maximum desired number of individuals (or other subject unit, such as families) who will complete the research Provide numbers for the site(s) reviewed by the UW IRB and for the study-wide total number; example: 20/100 |
|---|---|
| Design/Build: Senior Living Staff | 3 |
| Design/Build: Older Adults | 15 |
| Test: Senior Living or Senior Center Staff | 12 |
| Test: Older Adults | 120 |

**2.8 COVID-19 Screening**. If there will be any in-person interactions with the subjects, describe how you will screen them for COVID-19 symptoms within the 24 hours before the interaction. Also, describe the COVID-19 screening procedures for the study staff who will interact with the subjects.

Acceptable procedures include some type of symptom check or attestation, or a SARS-CoV-2 test with quick access to results. Symptom attestation involves an individual reviewing a list of symptoms and declaring the presence or absence of those symptoms. HSD strongly encourages adapting this Washington State Department of Health Screening Tool <a href="https://www.doh.wa.gov/Portals/1/Documents/1600/coronavirus/Employervisitorscreeningquidance.pdf">https://www.doh.wa.gov/Portals/1/Documents/1600/coronavirus/Employervisitorscreeningquidance.pdf</a> or the UW EH&S Example Symptom Self-Attestation in this document:

<u>https://www.ehs.washington.edu/system/files/resources/quidance-symptom-monitoring-COVID-19.pdf</u>. If you will test for the virus, you must also describe here whether the testing lab is CLIA-certified and how the results will be reported to the subjects.

Design/Build Phase: There will be no in-person interactions with subjects.

Test Phase: All assessments will take place remotely. The Stay Connected intervention is designed to be delivered via telephone. The control condition is a resource guide plus usual care for the senior living communities or senior centers which may include remote or in-person interactions but these will not be dictated by the study protocol.

# **3 NON-UW RESEARCH SETTING**

Complete this section only if UW investigators and people named in the <u>SUPPLEMENT:</u>
<u>Non-UW Individual Investigators</u> will conduct research procedures outside of UW and Harborview

**(3.1)**Reason for locations. Describe the reason(s) for choosing the locations.

This is especially important when the research will occur in locations or with populations that may be vulnerable to exploitation. One of the three ethical principles the IRB must consider is justice: ensuring that reasonable, non-exploitative, and well-considered procedures are administered fairly, with a fair distribution of costs and potential benefits.

We'll be working with 6 senior living communities or senior centers in the greater Seattle area.

**3.2**Local context. Culturally appropriate procedures and an understanding of local context are an important part of protecting subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect the research, how it is conducted, or how consent is obtained or documented.

Examples: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male researcher; instead, the researcher may need to ask a male family member for permission before the woman can be approached. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual members of a group. In some distinct cultural groups, signing forms may not be the norm.

This federal site maintains an international list of human research standards and requirements: <a href="http://www.hhs.gov/ohrp/international/index.html">http://www.hhs.gov/ohrp/international/index.html</a>

We will be recruiting locations both in and just outside of the greater Seattle Metro Area and do not anticipate any specific concerns with local context.

- **3.3** Location-specific laws. Describe any local laws that may affect the research (especially the research design and consent procedures). The most common examples are laws about:
  - **Specimens** for example, some countries will not allow biospecimens to be taken out of the country.
  - **Age of consent** laws about when an individual is considered old enough to be able to provide consent vary across states, and across countries.
  - **Legally authorized representative** laws about who can serve as a legally authorized representative (and who has priority when more than one person is available) vary across states and countries.
  - **Use of healthcare records** many states (including Washington State) have laws that are similar to the federal HIPAA law but that have additional requirements.

We do not anticipate any local laws that would affect research. Research data will be separate from healthcare records, and the study team will not have access to any healthcare records.

**3.4** Location-specific administrative or ethical requirements. Describe local administrative or ethical requirements that affect the research.

Example: A school district may require researchers to obtain permission from the head district office as well as school principals before approaching teachers or students; a factory in China may allow researchers to interview factory workers but not allow the workers to be paid for their participation.

We have received (and will receive for yet to be identified sites) permission from sites to recruit residents.

| 3.5 If the PI i | s a student: Does the research involve traveling outside of the US? |
|---|---|
| No | |
| Yes | → If yes, confirm by checking the box that (1) you will register with the <u>UW Office of Global Affairs</u> before traveling; (2) you will notify your advisor when the registration is complete; and (3) you will request a UW Travel Waiver if the research involves travel to the <u>list of countries</u> requiring a UW Travel Waiver. Confirmed |

# **4 RECRUITING and SCREENING PARTICIPANTS**

**4.1** Recruiting and Screening. Describe how subjects will be identified, recruited, and screened. Include information about: how, when, where, and in what setting. Identify who (by position or role, not name) will approach and recruit subjects, and who will screen them for eligibility.

#### Design/Build Phase

Senior Living Staff

- We will reach out to staff that participated in the survey phase (STUDY00010021) and gave us permission to contact them again in the future.

#### Older Adults

- We will reach out to older adults who, during the survey phase (STUDY00010021), indicated that they would be interested in working with the study team on future projects.

#### Test Phase

Senior Living or Senior Center Staff

- We will reach out to staff that have participated in previous phases of the study, and seek their assistance in identifying other participants.

#### Older Adults

- Older adults who are residents of senior living communities or members of senior centers will receive information about the study via flyers, newsletter postings, and ads. Staff at the senior living communities or senior centers may assist in distributing information about the study.
- Recruitment materials will encourage interested participants to contact the study team by email and/or phone. Please review uploaded examples of recruitment materials. Upon contact with the study team, the study team will complete an eligibility screening and obtain consent.

#### 4.2 Recruitment materials.

a. What materials (if any) will be used to recruit and screen subjects?

Examples: talking points for phone or in-person conversations; video or audio presentations; websites; social media messages; written materials such as letters, flyers for posting, brochures, or printed advertisements; questionnaires filled out by potential subjects.

## Design/Build Phase

For all participants (senior living staff and older adults) in this phase, we will email participants from the survey phase that gave us permission to contact them about participating in future phases of the project. We have uploaded examples of these recruitment emails to Zipline.

#### Test Phase

For senior living or senior center staff, we will work with participants from the Design/Build phase who express interest in continued work. For staff that have not participated in previous phases of the project, we will reach out to them by email.

For older adults, we will recruit older adults using flyers distributed by staff at the senior living communities or senior centers. We have uploaded examples of these flyers to Zipline.

We request flexibility/general approval of recruitment materials in order to have the ability to make minor changes to recruitment materials (i.e., changes that do not substantively alter the content of the project) without submitting a modification. We will submit modifications for changes that are more than minor.

**b.** Upload descriptions of each type of material (or the materials themselves) to **Zipline**. If letters or emails will be sent to any subjects, these should include a statement about how the subject's name and contact information were obtained. No sensitive information about the person (such as a diagnosis of a medical condition) should be included in the letter.

Version 2.50

HSD encourages researchers to consider uploading descriptions of most recruitment and screening materials instead of the materials themselves. The goal is to provide the researchers with the flexibility to change some information on the materials without submitting a Modification for IRB approval of the changes. Examples:

- Provide a list of talking points that will be used for phone or in-person conversations instead of a script.
- For the description of a flyer, include the information that it will provide the study phone number and the name of a study contact person (without providing the actual phone number or name). This means that a Modification would not be necessary if/when the study phone number or contact person changes. Also, instead of listing the inclusion/exclusion criteria, the description below might state that the flyer will list one or a few of the major inclusion/exclusion criteria.
- For the description of a video or a website, include a description of the possible visual elements and a list of the content (e.g., study phone number; study contact person; top three inclusion/exclusion criteria; payment of \$50; study name; UW researcher).

# **4.3** Relationship with participant population. Do any members of the study team have an existing relationship with the study population(s)?

Examples: a study team member may have a dual role with the study population (for example, being their clinical care provider, teacher, laboratory directory or tribal leader in addition to recruiting them for his/her research).



No Yes

→ If yes, describe the nature of the relationship.

#### **4.4 Payment to participants**. Describe any payment that will be provided, including:

- The total amount/value
- Whether payment will be "pro-rated" so that participants who are unable to complete the research may still receive some part of the payment

The IRB expects the consent process or study information provided to the subjects to include information about the number and amount of payments, and especially the time when subjects can expect to receive payment. One of the most frequent complaints received by HSD is from subjects who expected to receive cash or a check on the day that they completed a study and who were angry or disappointed when payment took 6-8 weeks to reach them.

Do not include a description of any expenses that will be reimbursed.

<u>Design/Build</u>: Each participant in this phase (both older adults and staff) will receive \$25 for their participation in co-design activities.

#### Test Phase

<u>Older Adult Participants</u>: Participants will complete 3 assessments (baseline, 4 weeks, and 9 weeks) and will receive \$15 for completing each of these assessments, for a total of \$45. We will offer participants either checks or Amazon gift codes as options for receiving these incentives.

Senior Living or Senior Center Staff: Participants will complete 2 assessments (baseline, 9 week) and will receive \$15 for completing each of these assessments, for a total of \$30. We will offer participants either checks or Amazon gift codes as options for receiving these incentives. Each senior living facility or senior center randomized to Stay Connected will receive \$3500 (to the facility not the individual) as incentive for staff time and administrative support.

| N/A | |
|---|---|
| 4.6 Will data or spe | ecimens be accessed or obtained for recruiting and screening procedures prior to enrollment? |
| - | and contact information; the information gathered from records that were screened; results of screening rescreening blood tests; Protected Health Information (PHI) from screening medical records to identify possible |
| | f no, skip the rest of this section; go to question 5.1. |
| I X I YAS | f yes, describe the data and/or specimens (including PHI) and whether it will be retained as part of the study data. |
| _ | Design/Build Phase Participants in this phase (both older adults and staff) provided consent during the survey phase (STUDY00010021) to be contacted about participating in future phases. Prior to consenting for the Design/Build phase, the potential participants will communicate with the study team by either phone or email. |
| | ruiting and screening. Will consent be obtained for any of the recruiting and screening |
| procedures? ( <u>Se</u> | ection 8: Consent of Adults asks about consent for the main study procedures). |
| | es: consent from individuals for their own participation; parental permission; assent from children; consent thorized representative for adult individuals who are unable to provide consent. |
| from the For a stu For a stu | ady in which names and contact information will be obtained from a registry: the registry should have consent a registry participants to release their names and contact information to researchers. Indy in which possible subjects are identified by screening records: there will be no consent process. Indy in which individuals respond to an announcement and call into a study phone line: the study team person to the individual may obtain non-written consent to ask eligibility questions over the phone. |
| _ | If no, skip the rest of this section; go to question <b>5.1</b> . |
| Yes → | If yes, describe the consent process. |
| • | <ul> <li>a. <u>Documentation of consent</u>. Will a written or verifiable electronic signature from the subject on a consent form be used to document consent for the <u>recruiting and screening procedures</u>?</li> <li>No If no, describe the information that will be provided during the consent process and for which procedures.</li> </ul> |
| | Yes → If yes, upload the consent form to <b>Zipline</b> . |
| | , . |

# **5 PROCEDURES**

**5.1 Study procedures**. Using lay language, provide a complete description of the study procedures, including the sequence, intervention or manipulation (if any), drug dosing information (if any), blood volumes and frequency of draws (if any), use of records, time required, and setting/location. If it is available: Upload a study flow sheet or table to **Zipline**.

For studies comparing standards of care: It is important to accurately identify the research procedures. See UW IRB POLICY:
Risks of Harm from Standard Care and the draft guidance from the federal Office of Human Research Protections, "Guidance on Disclosing Reasonably Foreseeable Risks in Research Evaluating Standards of Care"; October 20, 2014.

Information about pediatric blood volume and frequency of draws that would qualify for expedited review can be found in this reference table on the Seattle Children's IRB website.

## Design/Build Phase

Participants (both senior living community staff and older adults) will participate in user-centered design activities (e.g. focus groups, card sort activities, interviews) to co-design a supportive intervention modeled on Stay Connected, a menu-driven set of strategies to combat loneliness, anxiety and depression in older adults. We have uploaded a draft of an interview guide for initial use with older adults to provide information on topic areas that will be discussed as part of Design/Build activities. All study activities in this phase will take place remotely using technologies including Zoom (or other video conferencing technologies) and/or phone due to COVID-19 related restrictions.

#### **Test Phase**

Senior communities or senior centers will be randomized by community to receive either Stay Connected (as codesigned in the Design/Build phase) or a resource guide (e.g. Site A receives Stay Connected; Site B receives the resource guide). Staff at the senior living communities or senior centers will provide the intervention or the resource guide to enrolled participants. We have outlined the procedures for each participant group below.

Senior Living Community or Senior Center Staff/Intervention Deliverers After consent,

- 1. Staff will complete a brief demographics survey.
- 2. Staff who are randomized to the non-intervention group will receive a resource guide for both staff and residents consisting of virtual educational and entertainment opportunities, and stress and anxiety management tips. We have uploaded an example of the resource guide but request flexibility as we plan to update that resource guide with seasonal events and as ongoing opportunities become available.
- 3. Staff who are randomized to Stay Connected will complete a training on the Stay Connected intervention developed during the Design/Build phase of this project. We have uploaded a Stay Connected training manual
- 4. After training, both groups of staff will complete the following assessments of acceptability and usability (these measures have been uploaded to Zipline) either online using REDCap or by phone/videoconferencing (e.g. Zoom) with a study team member:
  - a. Acceptability of Intervention Measure (AIM)
  - b. Intervention Usability Scale (IUS)
  - c. Intervention Appropriateness Measure (IAM)
- 5. Staff delivering Stay Connected will deliver the intervention as developed in the design/build phase of this project. Stay Connected involves an initial assessment session followed by weekly calls for a total of 9 weeks of intervention. Please refer to the uploaded manual for more details.
- 6. Staff randomized to the resource guide will provide usual care to residents with the addition of a resource guide provided as needed by the staff to the older adults (at either the request of older adult for more resources or if the staff member assesses a need for additional resources as a need for the older adult).
- 7. 9 weeks after implementation of either Stay Connected or the resource guide, both groups of staff will complete the same measures of acceptability and usability:
  - a. Acceptability of Intervention Measures (AIM)

- b. Intervention Usability Scale (IUS)
- c. Intervention Appropriateness Measures (IAM)
- d. Stay Connected Provider Survey (uploaded to Zipline; previously used as part of STUDY00010527)

Members of the study team will complete fidelity reviews of Stay Connected sessions using the fidelity forms (uploaded to Zipline).

After the completion of the study, staff at senior living facilities or senior centers randomized to usual care will be offered the opportunity to receive training in Stay Connected.

#### Older Adult Participants

After consent,

- 1. Older adults will complete a baseline assessment prior to starting the intervention or receiving the resource guide. This assessment may be done either over the phone/videoconferencing (e.g. Zoom) with a member of the study team or online in REDCAP by the participant, depending on participant preference. The baseline assessment includes the following measures, which have been uploaded to Zipline as part of the survey phase:
  - a. Demographics,
  - b. Patient Health Questionnaire 9 Item (PHQ-9)
  - c. Generalized Anxiety Disorder 7 Item (GAD-7)
  - d. UCLA Loneliness Scale
  - e. Sheehan Disability Scale (SDS)
  - f. Behavioral Activation Scale (BADS)
  - g. PROMIS Social Isolation Short Version
- 2. After completion of baseline assessment, older adults will receive either the Stay Connected intervention for 9 weeks or the resource guide based on the randomization status of the community in which they reside or senior center they are a member of.
- 3. Follow Up Assessments: Older adult participants will complete follow up assessments 4 weeks and 9 weeks after starting Stay Connected or receiving the resource guide. These assessments may be done either over the phone with a member of the study team or online in REDCAP by the participant, depending on participant preference. The follow up assessments include the following measures:
  - a. Patient Health Questionnaire 9 Item (PHQ-9)
  - b. Generalized Anxiety Disorder 7 Item (GAD-7)
  - c. UCLA Loneliness Scale
  - d. Sheehan Disability Scale (SDS)
  - e. Behavioral Activation Scale (BADS)
  - f. PROMIS Social Isolation Short Version

Older adults in buildings or senior centers randomized to usual care will not be offered Stay Connected as part of the study. However, staff in those buildings or centers will be given the opportunity to be trained in Stay Connected to use in their buildings or centers after the study is complete.

| 5.2 Recording | gs. Does the research involve creating audio or video recordings? |
|---|---|
| No | → If no, go to <u>question <b>5.3</b>.</u> |
| X Yes | $\rightarrow$ If yes, verify that you have described what will be recorded in 5.1 and answer question <b>a</b> . |
| | a. Before recording, will consent for being recorded be obtained from subjects and any other<br>individuals who may be recorded? |
| | No |

| → If no, email <a href="mailto:hsdinfo@uw.edu">hsdinfo@uw.edu</a> before submitting this application in Zipline. In |
|---|
| the email, include a brief description of the research and a note that |
| individuals will be recorded without their advance consent. |



(5.3) MRI scans. Will any subjects have a Magnetic Resonance Imaging (MRI) scan as part of the study procedures?

This means scans that are performed solely for research purposes or clinical scans that are modified for research purposes (for example, using a gadolinium-based contrast agent when it is not required for clinical reasons).

| X | No |
|---|----|
| | Υe |

→ If no, go to question **5.4**.

es → If yes, answer questions a through c.

- a. Describe the MRI scan(s). Specifically:
  - What is the purpose of the scan(s)? Examples: obtain research data; safety assessment associated with a research procedure.
  - Which subjects will receive an MRI scan?
  - Describe the minimum and maximum number of scans per subject, and over what time period the scans will occur. For example: all subjects will undergo two MRI scans, six months apart.
- **b. Use of gadolinium**. Will any of the MRI scans involve the use of a gadolinium-based contrast agent (GBCA?)

| No |
|-----|
| Yes |

→ If yes, which agents will be used? Check all that apply.

| Brand Name | Generic Name | Chemical Structure |
|----------------------|--------------------------|--------------------|
| Dotarem | Gadoterate meglumine | Macrocylic |
| Eovist / Primovist | Gadoxetate disodium | Linear |
| Gadavist | Gadobutro | Macrocyclic |
| Magnevist | Gadpentetate dimeglumine | Linear |
| MultiHance | Gadobenate dimeglumine | Linear |
| Omniscan | Gadodiamide | Linear |
| OptiMARK | Gadoversetamide | Linear |
| ProHance | Gadoteridol | Macrocyclic |
| Other, provide name: | | |

1.) The FDA has concluded that gadolinium is retained in the body and brain for a significantly longer time than previously recognized, especially for linear GBCAs. The health-related risks of this longer retention are not yet clearly established. However, the UW IRB expects researchers to provide a compelling justification for using a linear GBCA instead of a macrocyclic GBCA, to manage the risks associated with GBCAs.

Describe why it is important to use a GBCA with the MRI scan(s). Describe the dose that will be used and (if it is more than the standard clinical dose recommended by the manufacturer) why it is necessary to use a higher dose. If a linear GBCA will be used, explain why a macrocyclic GBCA cannot be used.

2.) Information for subjects. Confirm by checking this box that subjects will be provided with the FDA-approved Patient Medication Guide for the GBCA being used in the research or that the same information will be inserted into the consent form.

Confirmed

c. MRI facility. At which facility(ies) will the MRI scans occur? Check all that apply.

UWMC Radiology/Imaging Services (the UWMC clinical facility)

DISC Diagnostic Imaging Sciences Center (UWMC research facility)

BMIC Biomolecular Imaging Center (South Lake Union research facility)

Harborview Radiology/Imaging Services (the Harborview clinical facility)

SCCA Imaging Services

Northwest Diagnostic Imaging

Other: identify in the text box below:

**Personnel.** For MRI scans that will be conducted at the DISC or BMIC research facilities: The role, qualifications, and training of individuals who will operate the scanner, administer the GBCA (if applicable), and/or insert and remove the IV catheter should be described in question **12.3**.

**5.4** Data variables. Describe the specific data that will be obtained (including a description of the most sensitive items). Alternatively, a list of the data variables may be uploaded to *Zipline*.

Design/Build: We have uploaded a draft of an interview guide to be used with older adults. Staff members will be interviewed about versions of the co-designed intervention and their impressions of the intervention, its acceptability, and ability to be implemented in their settings.

Test Phase

- Staff: Demographics, Acceptability of Intervention Measure (AIM), Intervention Usability Scale (IUS), Intervention Appropriateness Measure (IAM), Feasibility Intervention Measure (FIM), Stay Connected Provider Survey

- Older Adults: Demographics (including specifics on living arrangement), Patient Health Questionnaire 9 Item (PHQ-9), Generalized Anxiety Disorder 7 Item (GAD-7), UCLA Loneliness Scale, Sheehan Disability Scale (SDS), Behavioral Activation Scale (BADS), PROMIS Social Isolation
- (5.5) Data sources. For all types of data that will be accessed or collected for this research: Identify whether the data are being obtained from the subjects (or subjects' specimens) or whether they are being obtained from some other source (and identify the source).

If you have already provided this information in Question 5.1, you do not need to repeat the information here.

All data will be collected from subjects.

**5.6 Identifiability of data and specimens**. Answer these questions carefully and completely. This will allow HSD to accurately determine the type of review that is required and the relevant compliance requirements. Review the following definitions before answering the questions:

Access means to view or perceive data, but not to possess or record it. See, in contrast, the definition of "obtain".

Identifiable means that the identity of an individual is or may be readily (1) ascertained by the researcher or any other member of the study team from specific data variables or from a combination of data variables, or (2) associated with the information.

Direct identifiers are direct links between a subject and data/specimens. Examples include (but are not limited to): name, date of birth, medical record number, email or IP address, pathology or surgery accession number, student number, or a collection of data that is (when taken together) identifiable.

**Indirect identifiers** are information that links between direct identifiers and data/specimens. Examples: a subject code or pseudonym.

**Key** refers to a single place where direct identifiers and indirect identifiers are linked together so that, for example, coded data can be identified as relating to a specific person. Example: a master list that contains the data code and the identifiers linked to the codes.

**Obtain** means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. This is different from **accessing**, which means to view or perceive data.

| <b>a.</b> Will you or a | ny members of your team have <u>access</u> to any direct or indirect identifiers? |
|---|---|
| X Yes | → If yes, describe which identifiers and for which data/specimens. |
| | Names, Contact information (e.g. phone numbers, email addresses, mailing addresses) Date of Birth (older adult participants) |
| No | → If no, select the reason(s) why you (and all members of your team) will not have access to direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before access. |
| | There is an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to study team members under any circumstances. |
| | This agreement should be available upon request from the IRB. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |

| | There are other legal requirements prohibiting the release of the identifiers or key. Describe them below. |
|---|---|
| <b>b.</b> Will you or any | study team members obtain any direct or indirect identifiers? |
| X Yes | → If yes, describe which identifiers and for which data/specimens. |
| <u> </u> | Names, Contact information (e.g. phone numbers, email addresses, mailing addresses) Date of Birth (older adult participants) |
| No | → If no, select the reason(s) why you (and all members of your team) will not obtain direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before access. |
| | There will be an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) under any circumstances. |
| | This agreement should be available upon request from the IRB. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key. Describe them below. |
| • | rs will be obtained, indicate how the identifiers will be stored (and for which data). NOTE: Do e data security plan here – that information is requested in section 9.6. |
| | Identifiers will be stored with the data. Describe the data to which this applies: |
| | Identifiers and study data will be stored separately but a link will be maintained between the identifiers and the study data (for example, through the use of a code). Describe the data to which this applies: |
| | Names, Contact information (e.g. phone numbers, email addresses, mailing addresses) Date of Birth (older adult participants) |
| | Identifiers and study data will be stored separately, with no link between the identifiers and the study data. Describe the data to which this applies: |

| collaborator's institution/organization. |
|---|
| Examples include but are not limited to: (1) study, interpretation, or analysis of the data that results from the coded information or specimens; and (2) authorship on presentations or manuscripts related to this work. |
| No |
| <b>5.7</b> Protected Health Information (PHI). Will participants' identifiable PHI be accessed, obtained, used, or disclosed for any reason (for example, to identify or screen potential subjects, to obtain study data or specimens, for study follow-up) that does not involve the creation or obtaining of a Limited Data Set? |
| PHI is individually identifiable healthcare record information or clinical specimens from an organization considered a "covered entity" by federal HIPAA regulations, in any form or media, whether electronic, paper, or oral. You must answer yes to this question if the research involves identifiable health care records (e.g., medical, dental, pharmacy, nursing, billing, etc.), identifiable healthcare information from a clinical department repository, or observations or recordings of clinical interactions. |
| <b>X</b> No → If no, skip the rest of this question; go to question 5.8 |
| Yes → If yes, answer all of the questions below. |
| <b>a.</b> Describe the PHI and the reason for using it. Be specific. For example, will any "free text" fields (such as physician notes) be accessed, obtained, or used? |
| <b>b.</b> Is any of the PHI located in Washington State? |
| <ul> <li>No Yes</li> <li>c. Describe the pathway of how the PHI will be accessed or obtained, starting with the source/location and then describing the system/path/mechanism by which it will be identified, accessed, and copied for the research. Be specific. For example: directly view records; search through a department's clinical database; submit a request to Leaf.</li> </ul> |
| d. For which PHI will subjects provide HIPAA authorization before the PHI is accessed, obtained and/or used? |
| Confirm by checking the box that the UW Medicine HIPAA Authorization form maintained on the HSD website will be used to access, obtain, use, or disclose any UW Medicine PHI. |
| Confirmed |
| e. For which PHI will HIPAA authorization NOT be obtained from the subjects? |
| Provide the following assurances by checking the boxes. |
| The minimum necessary amount of PHI to accomplish the purposes described in this application will be accessed, obtained and/or used. |
| Document Date & Version Researcher Date & Version |
| 08/12/2020 03/11/2021 |

**d. Research collaboration**. Will individuals who provide coded information or specimens for the research also collaborate on other activities for this research? If yes, identify the activities and provide the name of the

Version 2.50

| The PHI will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study, or for other research for which the use or disclosure of PHI would be permitted. |
|---|
| The HIPAA "accounting for disclosures" requirement will be fulfilled, if applicable. See <a href="https://www.new.numer.com/"><u>UW</u></a> <a href="https://www.new.numer.com/">Medicine Compliance Policy #104</a> . |
| There will be reasonable safeguards to protect against identifying, directly or indirectly, any patient in any report of the research. |
| 5.8 Genomic data sharing. Will the research obtain or generate genomic data? |
| X No |
| Yes → If yes, answer the question below. |
| a. Will genomic data from this research be sent to a national database (for example, NIH's dbGaP database)? |
| No Yes → If yes, complete the <u>SUPPLEMENT Genomic Data Sharing</u> and upload it to <i>Zipline</i> . |
| 5.9 Whole genome sequencing. For research involving biospecimens: Will the research include whole genome sequencing? |
| Whole genome sequencing is sequencing of a human germline or somatic specimen with the intent to generate the genome or exome sequence of that specimen. |
| X No<br>Yes |
| 5.10 Possible secondary use or sharing of information, specimens, or subject contact information. Is it likely that the |
| <ul> <li>obtained or collected information, specimens, or subject contact information will be used for any of the following:</li> <li>Future research not described in this application (in other words, secondary research)</li> </ul> |
| <ul> <li>Submission to a repository, registry, or database managed by the study team, colleagues, or others for research purposes</li> </ul> |
| Sharing with others for their own research |
| Please consider the broadest possible future plans and whether consent will be obtained now from the subjects for future sharing or research uses (which it may not be possible to describe in detail at this time). Answer YES |
| even if future sharing or uses will use de-identified information or specimens. Answer <b>NO</b> if sharing is unlikely or if the only sharing will be through the NIH Genomic Data Sharing described in question 5.8. |
| Many federal grants and contracts now require data or specimen sharing as a condition of funding, and many journals require data sharing as a condition of publication. "Sharing" may include (for example): informal arrangements to share banked data/specimens with other investigators; establishing a repository that will formally share with other researchers through |

written agreements; or sending data/specimens to a third party repository/archive/entity such as the Social Science Open

Access Repository (SSOAR), or the UCLA Ethnomusicology Archive.

X Yes

- **Yes**  $\rightarrow$  If yes, answer all of the questions below.
  - **a.** Describe <u>what will be stored for future use</u>, including whether any direct or indirect (e.g., subject codes) identifiers will be stored.

All study data will be stored for future use. This includes all assessment (measures) data and needs assessment data. All data will be stored separately from identifiable information. Assessment data is coded with a unique study ID number, which cannot be used to identify the participant. The ID number will be stored along with the assessment data for future use.

**b.** Describe what will be shared with other researchers or with a repository/database/registry, including whether direct identifiers will be shared and (for specimens) what data will be released with the specimens.

All assessment data may be shared with other researchers. No direct identifiers will be shared. Participants consent to this sharing during the provision of informed consent.

c. Who will oversee and/or manage the sharing?

The oversight and/or management of the sharing will be the responsibility of the PI (Dr. Arean).

**d.** Describe the possible future uses, including limitations or restrictions (if any) on future uses or users. As stated above, consider the broadest possible uses.

Examples: data will be used only for cardiovascular research; data will not be used for research on population origins.

Possible future uses of this data include ongoing data analysis for publication and informing future grant proposals for clinical trials.

**e.** <u>Consent</u>. Will consent be obtained now from subjects for the secondary use, banking and/or future sharing?

No

Yes

- → If yes, be sure to include the information about this consent process in the consent form (if there is one) and in the answers to the consent questions in Section 8.
- **f.** Withdrawal. Will subjects be able to withdraw their data/specimens from secondary use, banking or sharing?

X No

Yes

→ If yes, describe how, and whether there are any limitations on withdrawal.

Example: data can be withdrawn from the repository but cannot be retrieved after they are released.

g. <u>Agreements for sharing or release</u>. Confirm by checking the box that the sharing or release will comply with UW (and, if applicable, UW Medicine) policies that require a formal agreement with the recipient for release of data or specimens to individuals or entities other than federal databases.

Data Use Agreements or Gatekeeping forms are used for data; Material Transfer Agreements are used for specimens (or specimens plus data). Do not attach any template agreement forms; the IRB neither reviews nor approves them

X Confirmed

**5.11 Communication with subjects during the study**. Describe the types of communication (if any) the research team will have with already-enrolled subjects during the study. Provide a description instead of the actual materials themselves.

Examples: email, texts, phone, or letter reminders about appointments or about returning study materials such as a questionnaire; requests to confirm contact information.

We may email or call participants to schedule appointments to complete surveys/questionnaires over the phone, remind participants to complete online surveys/questionnaires, and respond to questions about the study. We will also send gift codes or checks to participants via email or postal mail depending on participant preference.

**5.12 Future contact with subjects**. Is there a plan to retain any contact information for subjects so that they can be contacted in the future?



→ If yes, describe the purpose of the future contact, and whether use of the contact information will be limited to the study team; if not, describe who else could be provided with the contact information. Describe the criteria for approving requests for the information.

Examples: inform subjects about other studies; ask subjects for additional information or medical record access that is not currently part of the study proposed in this application; obtain another sample.

We will ask participants about their interest in participating in other studies and will document that answer. Contact information will be limited to our study teams (ALACRITY Center and CREATIV Lab). Requests for access outside of those groups will be approved by the PIs.

**5.13 Alternatives to participation.** Are there any alternative procedures or treatments <u>that might be advantageous</u> to the subjects?

If there are no alternative procedures or treatments, select "No". Examples of advantageous alternatives: earning extra class credit in some time-equivalent way other than research participation; obtaining supportive care or a standard clinical treatment from a health care provider instead of participating in research with an experimental drug.



→ If yes, describe the alternatives.

- **5.14 Upload to** *Zipline* all data collection forms (if any) that will be directly used by or with the subjects, and any scripts/talking points that will be used to collect the data. Do not include data collection forms that will be used to abstract data from other sources (such as medical or academic records), or video recordings.
  - **Examples**: survey, questionnaires, subject logs or diaries, focus group questions.
  - **NOTE:** Sometimes the IRB can approve the general content of surveys and other data collection instruments rather than the specific form itself. This prevents the need to submit a modification request for future minor changes that do not add new topics or increase the sensitivity of the questions. To request this general approval, use the text box below to identify the questionnaires/surveys/ etc. for which you are seeking this more general approval. Then briefly describe the scope of the topics that will be covered and the most personal and sensitive questions. The HSD staff person who screens this application will let you know whether this is sufficient or whether you will need to provide more information.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

For data that will be gathered in an evolving way: This refers to data collection/questions that are not pre-determined but rather are shaped during interactions with participants in response to observations and responses made during those interactions. If this applies to the proposed research, provide a description of the process by which the data collection/questions will be established during the interactions with subjects, how the data collection/questions will be documented, the topics likely to be addressed, the most sensitive type of information likely to be gathered, and the limitations (if any) on topics that will be raised or pursued.

## Use this text box (if desired) to provide:

- Short written descriptions of materials that cannot be uploaded, such as URLs
- A description of the process that will be used for data that will be gathered in an evolving way.
- The general content of questionnaires, surveys and similar instruments for which general approval is being sought. (See the **NOTE** bullet point in the instructions above.)

<u>Design/Build</u>: We request flexibility in data collection forms for this phase of the project as this phase is an interative, co-design process. We have uploaded an example draft of an interview guide for initial conversations with older adults. Staff members will be interviewed about versions of the co-designed intervention and their impressions of the intervention, its acceptability, and ability to be implemented in their settings.

Test Phase: All data collection forms have been uploaded to Zipline. Data will be collected by either REDCap or on the phone/videoconferencing (e.g., Zoom) based on participant preference.

5.15)SARS-CoV-2 testing. Will the subjects be tested for the SARS-CoV-2 coronavirus?

If the only testing is to screen the subjects (question 2.8), you do not need to answer this question



#### $\rightarrow$ If yes:

- Name the testing lab
- Confirm that the lab and its use of this test is CLIA-certified or certified by the Washington State Department of Health
- Describe whether you will return the results to the participants and, if yes, who will do it and how (including any information you would provide to subjects with positive test results).

5.16) Research equipment and COVID-19. Does you research involve any equipment that will be used on more than one subject that is not part of a clinical facility?

Examples: a computer tablet, a portable research ultra-sound device).



→ If yes: confirm by checking the box below that the disinfection and cleaning of the equipment will meet the enhanced UW Environmental Health & Safety requirements described here: https://www.ehs.washington.edu/system/files/resources/cleaning-disinfection-protocols-covid-19.pdf

Confirmed

# **6 CHILDREN (MINORS) and PARENTAL PERMISSION**

**6.1** Involvement of minors. Does the research include minors (children)?

**Minor or child** means someone who has not yet attained the legal age for consent for the research procedures, as described in the applicable laws of the jurisdiction in which the research will be conducted. This may or may not be the same as the definition used by funding agencies such as the National Institutes of Health.

- In Washington State the generic age of consent is 18, meaning that anyone under the age of 18 is considered a child.
- There are some procedures for which the age of consent is much lower in Washington State.

| | <ul> <li>The generic age of consent may be different in other states, and in other countries.</li> </ul> | | | | | |
|---|---|---|---|---|---|---|
| | <b>X</b> No $\rightarrow$ If no, go to Section 8. | | | | | |
| | Yes | → If yes, provide the age range the study population(s). If the | | | ge for cons | ent in |
| | Don't | <b>know</b> for some research in | volving social media | e age of the subjects. For examp<br>a, the Internet, or a dataset that<br>nt agency. Go to <u>Section 8</u> . | | - |
| s<br>p<br>re | ame as "pa<br>participate<br>eturned a | rmission. Parental permission massive" or "opt out" permission we because they have been provided orm indicating they don't want to be a later and face. | where it is assumed d with information | that parents are allowing their or<br>about the research and have no | children to | |
| а | . Will pare | ntal permission be obtained for: | | | | |
| | All of | the research procedures | → Go to <u>question</u> | <u> 6.2b.</u> | | |
| | None | of the research procedures | → Use the table<br>6.2b. | below to provide justification, a | nd skip qu | estion |
| | Some | of the research procedures | | below to identify the procedure ission will not be obtained. | es for whicl | 'n |
| | | nsider all research procedures and p<br>r future work. | plans, including screer | ing, future contact, and sharing/bo | anking of da | ta and |
| | Children<br>Group <sup>1</sup> | Describe the proce<br>data/specimen collecti<br>which there will be N<br>permission | on (if any) for<br>NO parental | Reason why parental permission will not be obtained | Will par<br>informe<br>the reso | d about |
| | | | | | | <b>_</b> |

Document Date & Version

Researcher Date & Version

| | <del></del> | <del></del> |
|---|---|---|
| Table footnotes | | |
| <ol> <li>If the answer is the same for all children groups or all procedures: collapse the answer across the groups ar</li> <li>If identifiable information or biospecimens will be obtained without parent permission, any waiver granted override parents' refusal to provide broad consent (for example, through the Northwest Biotrust).</li> <li>Will parents be informed about the research beforehand even though active permission is not being obtain</li> </ol> | by the IRB | |
| <b>b.</b> Indicate the plan for obtaining parental permission. One or both boxes must be checked. | | |
| Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably a only one parent has legal responsibility for the care and custody of the child | vailable; c | or when |
| One parent, even if the other parent is alive, known, competent, reasonably available, and responsibility for the care and custody of the child. | d shares le | egal |
| This is all that is required for minimal risk research. | | |
| If both boxes are checked, explain: | | |
| <b>6.3 Children who are wards.</b> Will any of the children be wards of the State or any other agency, insti | tution, or | entity? |
| Yes If yes, an advocate may need to be appointed for each child who is a ward. The adaddition to any other individual acting on behalf of the child as guardian or in loco same individual can serve as advocate for all children who are wards. | | |
| Describe who will be the advocate(s). The description must address the following | g points: | |
| <ul> <li>Background and experience</li> <li>Willingness to act in the best interests of the child for the duration of the</li> </ul> | e research | |
| <ul> <li>Independence of the research, research team, and any guardian organization</li> </ul> | ation | |
| 7 ASSENT OF CHILDREN (MINORS) | | |
| Go to <u>Section 8</u> if your research does not involve children (minors). | | |
| <b>7.1 Assent of children (minors)</b> . Though children do not have the legal capacity to "consent" to particle research, they should be involved in the process if they are able to "assent" by having a study expand/or by reading a simple form about the study, and then giving their verbal choice about wheth participate. They may also provide a written assent if they are older. See <a href="WORKSHEET Children">WORKSHEET Children</a> in which a child's assent may be unnecessary or inappropriate. | plained to<br>her they v | vant to |
| a. Will assent be obtained for: | | |
| All research procedures and child groups → Go to question 7.2. | | |

| | None of the resea | arch procedures and child groups | → Use the table below to provide justification,<br>then skip to <u>question 7.6</u> |
|---|---|---|---|
| | Some of your rese | earch procedures and child groups | Use the table below to identify the procedures for which assent will not be obtained. |
| | to consider all rese<br>ns for future work. | arch procedures and plans, including scree | ning, future contact, and sharing/banking of data and |
| Child | ren Group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which assent will NOT be obtained | Reason why assent will not be obtained |
| Table footn 1. If the an | | or all children groups or all procedures, col | lapse your answer across the groups and/or procedures. |
| differer | it ages, answer se | | n child group. If the research involves children of n are non-English speakers, include a description of . |
| | | escribe how a child's objection or resis ified during the research, and what th | tance to participation (including non-verbal e response will be. |
| | • | • | tronic signatures, etc.) be used to present assent atures) of assent? If yes, describe how this will be |
| <b>7.5 Docume</b> obtaine | | t. Which of the following statements | describes whether documentation of assent will be |
| No | ne of the researd | ch procedures and child groups | → Use the table below to provide justification, then go to <u>question <b>7.5.b</b></u> |
| All | of the research p | procedures and child groups | → Go to <u>question <b>7.5.a</b></u> , do not complete the table |
| So | me of the researd | ch procedures and/or child groups | |
| Document Da | te & Version | | Researcher Date & Version |

→ Complete the table below and then to go question 7.5.a Describe the procedures or data/specimen collection (if any) for which assent Children Group<sup>1</sup> will NOT be documented Table footnotes 1. If the answer is the same for all children groups or all procedures, collapse the answer across the groups and/or procedures. a. Describe how assent will be documented. If the children are functionally illiterate or are not fluent in English, include a description of the documentation process for them. b. Upload all assent materials (talking points, videos, forms, etc.) to Zipline. Assent materials are not required to provide all of the standard elements of adult consent; the information should be appropriate to the age, population, and research procedures. The documents should be in Word, if possible. 7.6 Children who reach the legal age of consent during participation in longitudinal research. Children who were enrolled at a young age and continue for many years: It is best practice to re-obtain assent (or to obtain it for the first time, if it was not obtained at the beginning of their participation). Children who reach the legal age of consent: Informed consent must be obtained from the now-adult subject for (1) any ongoing interactions or interventions with the subjects, or (2) the continued analysis of specimens or data for which the subject's identify is readily identifiable to the researcher, unless the IRB waives this requirement. **a.** Describe the plans (if any) to re-obtain assent from children. **b.** Describe the plans (if any) to obtain consent for children who reach the legal age of consent. If adult consent will be obtained from them, describe what will happen regarding now-adult subjects who cannot be contacted. If consent will not obtained or will not be possible: explain why. 7.7 Other regulatory requirements. (This is for information only; no answer or response is required.) Researchers are

7.7 Other regulatory requirements. (This is for information only; no answer or response is required.) Researchers are responsible for determining whether their research conducted in schools, with student records, or over the Internet comply with permission, consent, and inspection requirements of the following federal regulations:

- PPRA Protection of Pupil Rights Amendment
- FERPA Family Education Rights and Privacy Act
- COPPA Children's Online Privacy Protection Act

# **8 CONSENT OF ADULTS** Review the following definitions before answering the questions in this section. is the process of informing potential subjects about the research and asking them whether they want to participate. It does not necessarily include the signing of a CONSENT consent form. refers to how a subject's decision to participate in the research is documented. CONSENT DOCUMENTATION This is typically obtained by having the subject sign a consent form. is a document signed by subjects, by which they agree to participate in the **CONSENT FORM** research as described in the consent form and in the consent process. **ELEMENTS OF CONSENT** are specific information that is required to be provided to subjects. are the qualities of the consent process as a whole. These are: Consent must be legally effective. The process minimizes the possibility of coercion or undue influence. Subjects or their representatives must be given sufficient opportunity to discuss and consider participation.

**CHARACTERISTICS OF CONSENT** 

- The information provided must:
  - Begin with presentation of key information (for consent materials over 2,000 words)
  - Be what a reasonable person would want to have
  - Be organized and presented so as to facilitate understanding
  - Be provided in sufficient detail
  - Not ask or appear to ask subjects to waive their rights

#### is the parent's active permission for the child to participate in the research. PARENTAL PERMISSION Parental permission is subject to the same requirements as consent, including written documentation of permission and required elements.

# **SHORT FORM CONSENT**

is an alternative way of obtaining written documentation of consent that is most commonly used with individuals who are illiterate or whose language is one for which translated consent forms are not available.

means there is IRB approval for not obtaining consent or for not including some of the elements of consent in the consent process.

#### **WAIVER OF CONSENT**

**NOTE**: If you plan to obtain identifiable information or identifiable biospecimens without consent, any waiver granted by the IRB does not override a subject's refusal to provide broad consent (for example, the Northwest Biotrust).

## WAIVER OF DOCUMENTATION OF CONSENT

means that there is IRB approval for not obtaining written documentation of

**8.1 Groups** Identify the groups to which the answers in this section apply.

Adult subjects

| | <b>a</b> . Are ther | e any procedures for which consent will no | ot be obtained? | | |
|---|---|---|---|---|---|
| | X No<br>Yes | → If yes, use the table below to identify is an acceptable answer for some study | the procedures for which consent will not<br>dies. | : be obtaine | ed. "All" |
| | Be sure to cor future work. | nsider all research procedures and plans, includ | ding future contact, and sharing/banking of da | nta and speci | imens for |
| | Group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which there will be NO consent process | Reason why consent will not be obtained | Will subj<br>provide<br>info abo<br>researc<br>they fi<br>YES | ed with<br>out the<br>h after |
| <u>Tai</u><br>1. | | r is the same for all groups, collapse your answe | | !! arounc | |
| | | the consent process, if consent will be obtagroups and procedures separately if the con | • | all groups. | |
| | <ul><li>Who</li><li>How</li><li>part</li></ul> | o include: location/setting where consent will be obtaine o will obtain consent (refer to positions, roles, o v subjects will be provided sufficient opportunit ticipation t/assent will be obtained via the modality (p | or titles, not names)<br>ty to discuss the study with the research team ( | | r |

APPLICATION IRB Protocol

Researcher Date & Version

03/11/2021

Version 3.1 Page 33 of 51

Parents who are providing permission for their children to participate in research

procedures except recruiting and screening and, if yes, how.

to question 4.6.

Document Date & Version

08/12/2020

Version 2.50

permission and "subjects" should also be interpreted as applying to the parents.

→ If you selected **PARENTS**, the word "consent" below should also be interpreted as applying to parental

8.2 The consent process and characteristics. This series of questions is about whether consent will be obtained for all

The issue of consent for recruiting and screening activities is addressed in question 4.7. You do not need to repeat your answer

#### Design/Build Phase

Participants in this phase will be recruited from study phase participants that gave permission for the study team to contact them about participating in future work. We will contact the participants by email with information about the design/build phase and invite those interested to contact the study team by phone or email. If participants did not provide an email during the survey phase, we will contact those individuals by phone. We will either email the consent form to participants or review it on the phone with participants. All participants will have access to a study team member by phone and/or email to answer questions. Consent will be documented by the study team in REDCap. The consent form has been uploaded to Zipline.

# Test Phase

Senior living community or senior center staff will be consented for this phase by phone or email prior to the training on the intervention that they are randomized to. We will email a link to a REDCap survey that has the consent form and demographics. If a participant prefers to complete the consent and demographics survey over the phone, a study team member will do that. Participants will have the chance to ask questions of the study team by email or phone. The consent form has been uploaded to Zipline.

Older Adults will be consented prior to completion of the baseline assessments. If a participant has chosen to complete the baseline assessment on the phone with a study team member, they will complete the consent on the phone. If the participant choses to complete the baseline assessment online, they will review and complete the consent in REDCap. The consent form has been uploaded to Zipline.

**c.** <u>Comprehension</u>. Describe the methods that will be used to ensure or test the subjects' understanding of the information during the consent process.

## Design/Build

Participants will have the opportunity to ask questions of study staff and, prior to starting co-design activities, study staff will review procedures and provide additional opportunities to ask questions.

#### **Test Phase**

Participants will have the opportunity to ask questions of study staff at all times.

If an older adult participant choses to complete the consent and baseline assessment online, they will be asked to complete the following consent quiz to ensure comprehension:

Being in the research study is voluntary. TRUE/FALSE

True: That's right! Being in this study is completely voluntary and you can stop at any time. False: Good try! Actually, being in this study is voluntary and you can stop at any time.

No one other than the people working on the study will see my answers to the questions, unless I may be in an unsafe situation. TRUE/FALSE

True: That's right! We will kept all of your answers private. The only time that we would need to tell someone else is if we are concerned about your safety.

False: Nice try! We actually do keep all of your answers private. The only time that we would need to tell someone else is if we are concerned about your safety.

If the participant is completing consent procedures over the phone, study team members will prompt for questions and understanding prior to seeking consent.

Version 2.50

**d.** <u>Influence</u>. Does the research involve any subject groups that might find it difficult to say "no" to participation because of the setting or their relationship with someone on the study team, even if they aren't pressured to participate?

Examples: Student participants being recruited into their teacher's research; patients being recruited into their healthcare provider's research, study team members who are participants; outpatients recruited from an outpatient surgery waiting room just prior to their surgery.

| Χ | No |
|---|-----|
| | Yes |

→ If yes, describe what will be done to reduce any effect of the setting or relationship on the participation decision.

Examples: a study coordinator will obtain consent instead of the subjects' physician; the researcher will not know which subjects agreed to participate; subjects will have two days to decide after hearing about the study.

e. Information provided is tailored to needs of subject population. Describe the basis for concluding that the information that will be provided to subjects (via written or oral methods) is what a reasonable member of the subject population(s) would want to know. If the research consent materials contain a key information section, also describe the basis for concluding that the information presented in that section is that which is most likely to assist the selected subject population with making a decision. See GUIDANCE Key Information for Consent Materials.

For example: Consultation with publications about research subjects' preferences, disease-focused nonprofit groups, patient interest groups, or other researchers/study staff with experience with the specific population. It may also involve directly consulting selected members of the study population.

Our team has extensive experience working with older adults, including those experiencing depression, anxiety, loneliness, etc; co-design of psychosocial interventions; and remote research. The consent methods outlined here are modeled on previous work by the PIs of this project.

**f.** Ongoing process. For research that involves multiple or continued interaction with subjects over time, describe the opportunities (if any) that will be given to subjects to ask questions or to change their minds about participating.

<u>Design/Build</u>: We anticipate that we may interact with participants a couple of times during this iterative, codesign process. Prior to each interaction, study staff will review procedures, allow time for questions, and allow participants the opportunity to change their minds about participating.

<u>Test</u>: Study staff will interact with participants for follow-up assessments at Weeks 4 and 9. During these interactions, study staff will review procedures, allow time for questions, and allow participants the opportunity to change their minds about participating.

**8.3 Electronic presentation of consent information.** Will any part of the consent-related information be provided electronically for some or all of the subjects?

This refers to the use of electronic systems and processes instead of (or in addition to) a paper consent form. For example, an emailed consent form, a passive or an interactive website, graphics, audio, video podcasts. See <u>GUIDANCE Electronic Informed Consent</u> for information about electronic consent requirements at UW.



→ If no, skip to <u>question 8.4</u>
## Yes → If yes, answer questions a through e

a. Describe the electronic consent methodology and the information that will be provided.

All informational materials must be made available to the IRB. Website content should be provided as a Word document. It is considered best practice to give subjects information about multi-page/multi-screen information that will help them assess how long it will take them to complete the process. For example, telling them that it will take about 15 minutes, or that it involves reading six screens or pages.

This is detailed in 8.2b and 8.2c.

**b.** Describe how the information can be navigated (if relevant). For example, will the subject be able to proceed forward or backward within the system, or to stop and continue at a later time?

The participant will review the consent information on a website from REDCap. The participant may leave the consent form and return at a later date, but their progress would not be saved.

c. In a standard paper-based consent process, the subjects generally have the opportunity to go through the consent form with study staff and/or to ask study staff about any question they may have after reading the consent form. Describe what will be done, if anything, to facilitate the subject's comprehension and opportunity to ask questions when consent information is presented electronically. Include a description of any provisions to help ensure privacy and confidentiality during this process.

Examples: hyperlinks, help text, telephone calls, text messages or other type of electronic messaging, video conference, live chat with remotely located study team members.

Contact information for the study team is provided. Additionally, participants will be asked to answer a Yes/No question of "Do you have any questions?" If the participant answers Yes, the participant will be prompted to contact the study team member and will be alerted a member of the study team will contact them if we haven't heard from them. The consent form and all fields completed by the participant populate a REDCap database, which ensures privacy and confidentiality of responses.

d. What will happen if there are individuals who wish to participate but who do not have access to the consent methodology being used, or who do not wish to use it? Are there alternative ways in which they can obtain the information, or will there be some assistance available? If this is a clinical trial, these individuals cannot be excluded from the research unless there is a compelling rationale.

For example, consider individuals who lack familiarity with electronic systems, have poor eyesight or impaired motor skills, or who do not have easy email or internet access.

Participants will be given the option to complete study procedures, including consent, online or by phone.

**e**. How will additional information be provided to subjects during the research, including any significant new findings (such as new risk information) If this is not an issue, explain why.

If necessary, we will contact participants via the modality that they selected to complete study procedures (phone or email).

**8.4 Written documentation of consent.** Which of the statements below describe whether documentation of consent will be obtained? NOTE: This question does not apply to screening and recruiting procedures which have already been addressed in <u>question 4.7</u>.

Documentation of consent that is obtained electronically is not considered written consent unless it is obtained by a method that allows verification of the individual's signature. In other words, saying "yes" by email is rarely considered to be written documentation of consent

| a. Is written documentation of consent being obtained for: | | | | |
|---|---|---|---|---|
| X None of the research procedures | | → Use the table below to provide justification th<br>8.5. | | |
| All of | the research procedures | → Do not complete the table; go to question <b>8.4</b> | <u>.b.</u> | |
| Some | of the research procedures | → Use the table below to identify the procedure<br>documentation of consent will not be obtaine<br>subjects. | | |
| Adult<br>subject<br>group <sup>1</sup> | | data/specimen collection (if any) for which NO documentation of consent | Will the provided write states described research (option YES | with a ten ment ing the arch |
| Older Adults | consent will be documented in I | e methods described in 8.2b and 8.2c. Provision of REDCap either automatically upon completion of the study team if completing consent procedures | х | |
| Senior Living<br>Community or<br>Senior Center<br>Staff | Consent will be obtained via the consent will be documented in I consent procedures online or by | e methods described in 8.2b and 8.2c. Provision of REDCap either automatically upon completion of the study team if completing consent procedures | x | |

#### Table footnotes

1. If the answer is the same for all adult groups or all procedures, collapse the answer across the groups and/or procedures.

| No Yes If yes, describe the methodology that will be used. See the GUIDANCE Electronic Informed Consent for information about options (including the DocuSign system available through UW-IT) and requirements. D.1 is this method legally valid in the jurisdiction where the research will occur? | • | FDA-regulated studies must use a system that complies with the FDA's "Part 11" requirements about electronic systems and records. Note that the UW-IT supported DocuSign e-signature system does not meet this requirement. Having subjects check a box at the beginning of an emailed or web-based questionnaire is not considered legally effective documentation of consent. |
|---|---|---|
| See the GUIDANCE Electronic Informed Consent for information about options (including the DocuSign system available through UW-IT) and requirements. b.1 is this method legally valid in the jurisdiction where the research will occur? No | | No |
| b.2 Will verification of the subject's identity be obtained if the signature is not personally witnessed by a member of the study team? Note that this is required for FDA-regulated studies. See the GUIDANCE Electronic Informed Consent for information and examples No If no, provide the rationale for why this is appropriate. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consent signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcats to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | See the <u>GUIDANCE Electronic Informed Consent</u> for information about options (including the DocuSign |
| b.2 Will verification of the subject's identity be obtained if the signature is not personally witnessed by a member of the study team? Note that this is required for FDA-regulated studies. See the GUIDANCE Electronic Informed Consent for information and examples No If no, provide the rationale for why this is appropriate. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consent signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcats to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | |
| b.2 Will verification of the subject's identity be obtained if the signature is not personally witnessed by a member of the study team? Note that this is required for FDA-regulated studies. See the GUIDANCE Electronic Informed Consent for information and examples No → If no, provide the rationale for why this is appropriate. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consent signature? Yes → If yes, how? b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | <b>b.1</b> Is this method legally valid in the jurisdiction where the research will occur? |
| witnessed by a member of the study team? Note that this is required for FDA-regulated studies. See the GUIDANCE Electronic Informed Consent for information and examples No If no, provide the rationale for why this is appropriate. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consent signature? Yes If yes, how? b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | $oldsymbol{arphi}$ |
| witnessed by a member of the study team? Note that this is required for FDA-regulated studies. See the GUIDANCE Electronic Informed Consent for information and examples No If no, provide the rationale for why this is appropriate. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consent signature? Yes If yes, how? b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | |
| No | | witnessed by a member of the study team? Note that this is required for FDA-regulated |
| be the risks to the actual subject if somebody other than the intended signer provides the consent signature? Yes If yes, how? b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | See the <b>GUIDANCE Electronic Informed Consent</b> for information and examples |
| b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | be the risks to the actual subject if somebody other than the intended |
| b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | signer provides the consent signature. |
| b.3 How will the requirement be met to provide a copy of the consent information (consent form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | Yes →If yes, how? |
| form) to individuals who provide an e-signature? The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | |
| email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. 8.5 Non-English-speaking or -reading adult subjects. Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? | | |
| or who lack fluency or literacy in English? | | email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration |
| or who lack fluency or literacy in English? | | |
| X No | XN | o |
| Document Date & Version Researcher Date & Version | Document Da | ate & Version Researcher Date & Version |

b. Electronic consent signature. For studies in which documentation of consent will be obtained: will subjects use

an electronic method to provide their consent signature?

| <u></u> | If yes, describe the process that will be used to ensure that the oral and written information provided to them during the consent process and throughout the study will be in a language readily understandable to them and (for written materials such as consent forms or questionnaires) at an appropriate reading/comprehension level. |
|---|---|
| | a. <u>Interpretation</u> . Describe how interpretation will be provided, and when. Also, describe the qualifications of the interpreter(s) – for example, background, experience, language proficiency in English and in the other language, certification, other credentials, familiarity with the research-related vocabulary in English and the target language. |
| | <b>b.</b> <u>Translations</u> . Describe how translations will be obtained for all study materials (not just consent forms). Also, describe the method for ensuring that the translations meet the UW IRB's requirement that translated documents will be linguistically accurate, at an appropriate reading level for the participant population, and culturally sensitive for the locale in which they will be used. |
| documentation | tten documentation of consent. There are many possible barriers to obtaining written of consent. Consider, for example, individuals who are functionally illiterate; do not read English ensory or motor impairments that may impede the ability to read and sign a consent form. |
| have difficul | plans (if any) for obtaining written documentation of consent from potential subjects who may ty with the standard documentation process (that is, reading and signing a consent form). Skip this written documentation of consent is not being obtained for any part of the research. |
| | solutions: Translated consent forms; use of the Short Form consent process; reading the form to the person ign it; excluding individuals who cannot read and understand the consent form. |
| N/A | |
| Note: "Blinding" time that they w X No Yes | I information be deliberately withheld, or will false information be provided, to any of the subjects? subjects to their study group/condition/arm is not considered to be deception, but not telling them ahead of will be subject to an intervention or about the purpose of the procedure(s) is deception. If yes, describe what information and why. |
| [ | Example: It may be necessary to deceive subjects about the purpose of the study (describe why). |

| <ul> <li>a. Will subjects be informed beforehand that they will be unaware of or misled regarding the nature or purposes of the research? (Note: this is not necessarily required.)</li> <li>No</li> <li>Yes</li> </ul> | |
|---|---|
| <b>b.</b> Will subjects be debriefed later? (Note: this is not necessarily required.) | |
| No Yes → If yes, describe how and when this will occur. Upload any debriefing materials, including talking points or a script, to <b>Zipline</b> . | |
| .8 Cognitively impaired adults, and other adults unable to consent. Will such individuals be included in the | |
| research? Examples: individuals with Traumatic Brain Injury (TBI) or dementia; individuals who are unconscious, or who are significantly intoxicated. | / |
| <b>X</b> No $\rightarrow$ If no, go to <u>question 8.9</u> . | |
| Yes → If yes, answer the following questions. | |
| a. Rationale. Provide the rationale for including this population. | |
| <b>b.</b> Capacity for consent / decision making capacity. Describe the process that will be used to | |
| determine whether a cognitively impaired individual is capable of consent decision making with respect to the research protocol and setting. | |
| <b>b.1.</b> If there will be repeated interactions with the impaired subjects over a time period whe cognitive capacity could increase or diminish, also describe how (if at all) decision-making capacity will be re-assessed and (if appropriate) consent obtained during that time. | n |
| c. <u>Permission (surrogate consent)</u> . If the research will include adults who cannot consent for<br>themselves, describe the process for obtaining permission ("surrogate consent") from a legall<br>authorized representative (LAR). | ly |
| For research conducted in Washington State, see the <b>GUIDANCE Legally Authorized Representative</b> to learn which individuals meet the state definition of "legally authorized representative". | |

| | d. <u>Assent</u> . Describe whether assent will be required of all, some, or none of the subjects. If some, indicate which subjects will be required to assent and which will not (and why not). Describe any process that will be used to obtain and document assent from the subjects. |
|---|---|
| | <b>e.</b> <u>Dissent or resistance</u> . Describe how a subject's objection or resistance to participation (including non-verbal) during the research will be identified, and what will occur in response. |
| 8.9 Re | esearch use of human fetal tissue obtained from elective abortion. Federal and UW Policy specify some |
| | quirements for the consent process. If you are conducting this type of research, check the boxes to confirm |
| th | ese requirements will be followed. |
| | Informed consent for the donation of fetal tissue for research use will be obtained by someone other than |
| | the person who obtained the informed consent for abortion. |
| | Informed consent for the donation of fetal tissue for research use will be obtained after the informed consent for abortion. |
| | Participation in the research will not affect the method of abortion. |
| | No enticements, benefits, or financial incentives will be used at any level of the process to incentivize |
| | abortion or the donation of human fetal tissue. |
| | The informed consent form for the donation of fetal tissue for use in research will be signed by both the |
| | woman and the person who obtains the informed consent. |
| 0 10 0 | Concept related materials. Unload to <b>Zipling</b> all concept carints /talking points, concept forms, debriofing |

- **8.10 Consent-related materials**. Upload to *Zipline* all consent scripts/talking points, consent forms, debriefing statements, Information Statements, Short Form consent forms, parental permission forms, and any other consent-related materials that will be used. Materials that will be used by a specific site should be uploaded to that site's **Local Site Documents** page.
  - <u>Translations must be submitted and approved before they can be used</u>. However, we strongly encourage you to wait to provide them until the IRB has approved the English versions.
  - <u>Combination forms</u>: It may be appropriate to combine parental permission with consent, if parents are subjects as well as providing permission for the participation of their children. Similarly, a consent form may be appropriately considered an assent form for older children.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. URLs (website addresses) may also be provided, or written descriptions of websites. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

### 9 PRIVACY AND CONFIDENTIALITY

**9.1 Privacy protections.** Describe the steps that will be taken, if any, to address possible privacy concerns of subjects and potential subjects.

Privacy refers to the sense of being in control of access that others have to ourselves. This can be an issue with respect to recruiting, consenting, sensitivity of the data being collected, and the method of data collection. Examples:

- Many subjects will feel a violation of privacy if they receive a letter asking them to participate in a study because they
  have \_\_\_\_ medical condition, when their name, contact information, and medical condition were drawn from medical
  records without their consent. Example: the IRB expects that "cold call" recruitment letters will inform the subject
  about how their information was obtained.
- Recruiting subjects immediately prior to a sensitive or invasive procedure (e.g., in an outpatient surgery waiting room) will feel like an invasion of privacy to some individuals.
- Asking subjects about sensitive topics (e.g. details about sexual behavior) may feel like an invasion of privacy to some individuals.

We will be asking about the impact of stressful life events; we highlight in the consent that we will discuss these topics and let participants know that they are able to skip any questions they choose or withdraw from the study at any time.

| 9.2 | Iden | tification of individuals in publications and presentations. Will potentially identifiable information about |
|---|---|---|
| | subje | ects be used in publications and presentations, or is it possible that individual identities could be inferred from |
| | what | t is planned to be published or presented? |
| | X | No |
| | | <b>Yes</b> → If yes, will subject consent be obtained for this use? |

| If ye | s, will s | subject consent be obtained for this use? |
|---|---|---|
| | Yes | |
| | No | ightarrow If no, describe the steps that will be taken to protect subjects (or small groups of |
| | _ | subjects) from being identifiable. |

- 9.3 State mandatory reporting. Each state has reporting laws that require some types of individuals to report some kinds of abuse, and medical conditions that are under public health surveillance. These include:
  - Child abuse
  - Abuse, abandonment, neglect, or financial exploitation of a vulnerable adult
  - Sexual assault
  - Serious physical assault
  - Medical conditions subject to mandatory reporting (notification) for public health surveillance

Are you or a member of the research team likely to learn of any of the above events or circumstances while conducting the research **AND** feel obligated to report it to state authorities?

No X Yes

→ If yes, the UW IRB expects subjects to be informed of this possibility in the consent form or during the consent process, unless you provide a rationale for not doing so:

<u>Design/Build</u>: While unlikely given the nature of the interactions with participants, we do inform participants of this possibility in the assent/consent. Please refer to the uploaded consent/assent forms.

<u>Test Phase</u>: We inform participant of this possibility in the consent process. If study team members learn of any information that would require reporting, study staff will make appropriate reports.

If staff at senior living communities or senior centers learn of such information, they will make the report following procedures unique to their setting.

9.4 Retention of identifiers and data. Check the box below to indicate assurance that any identifiers (or links between identifiers and data/specimens) and data that are part of the research records will not be destroyed until after the end of the applicable records retention requirements (e.g. Washington State; funding agency or sponsor; Food and Drug Administration). If it is important to say something about destruction of identifiers (or links to identifiers) in the consent form, state something like "the link between your identifier and the research data will be destroyed after the records retention period required by state and/or federal law."

This question can be left blank for conversion applications (existing paper applications that are being "converted" into a Zipline application.)

See the "Research Data" sections of the following website for UW Records management for the Washington State research rectords retention schedules that apply in general to the UW (not involving UW Medicine data):

http://f2.washington.edu/fm/recmgt/gs/research?title=R

See the "Research Records and Data" information in Section 8 of this document for the retention schedules for UW Medicine Records: <a href="https://www.uwmedicine.org/recordsmanagementuwm-records-retention-schedule.pdf">https://www.uwmedicine.org/recordsmanagementuwm-records-retention-schedule.pdf</a>



- **9.5 Certificates of Confidentiality**. Will a federal Certificate of Confidentiality be obtained for the research data? *NOTE: Answer "No" if the study is funded by NIH or the CDC, because all NIH-funded and CDC-funded studies automatically have a Certificate.* 
  - X No Yes
- (9.6) Data and specimen security protections. Identify the data classifications and the security protections that will be provided for all sites where data will be collected, transmitted, or stored, referring to the GUIDANCE Data and Security Protections for the minimum requirements for each data classification level. It is not possible to answer this question without reading this document. Data security protections should not conflict with records retention requirements.
  - **a.** Which level of protections will be applied to the data and specimens? If more than one level will be used, describe which level will apply to which data and which specimens and at which sites.

Level 3

- **b.** Use this space to provide additional information, details, or to describe protections that do not fit into one of the levels. If there are any protections within the level listed in 9.6.a which will *not* be followed, list those here, including identifying the sites where this exception will apply.
  - Study data will be labeled with a unique study identification number. Only the relevant project staff will have access to the master list linking subject names to study identification numbers. The master list will be kept separate from the coded study data.
  - All identifying information collected as part of the study will be stored in a database on a secure server which is password protected with limited access by the study team.
  - Publications or presentation of findings will not include information identifying the subjects.

### 10 RISK / BENEFIT ASSESSMENT

- **10.1** Anticipated risks. Describe the <u>reasonably foreseeable</u> risks of harm, discomforts, and hazards to the subjects and others of the research procedures. For each harm, discomfort, or hazard:
  - Describe the magnitude, probability, duration, and/or reversibility of the harm, discomfort, or hazard, AND
  - Describe how the risks will be reduced or managed. Do not describe data security protections here, these are already described in Question 9.6.
  - Consider possible physical, psychological, social, legal, and economic harms, including possible negative effects on financial standing, employability, insurability, educational advancement or reputation. For example, a breach of confidentiality might have these effects.
  - Examples of "others": embryo, fetus, or nursing child; family members; a specific group.
  - Do not include the risks of non-research procedures that are already being performed.
  - If the study design specifies that subjects will be assigned to a specific condition or intervention, then the condition or intervention is a research procedure even if it is a standard of care.
  - Examples of mitigation strategies: inclusion/exclusion criteria; applying appropriate data security measures to prevent unauthorized access to individually identifiable data; coding data; taking blood samples to monitor something that indicates drug toxicity.
  - As with all questions on this application, you may refer to uploaded documents.

Subjects may experience emotional discomfort as a result of the topics discussed.

It is possible that in the course of our study procedures we determine that a report should be made for abuse of an elder, child, or dependent adult. In addition, we are mandated to report the abandonment, isolation, neglect, or financial abuse of an elder, child, or dependent adult; and/or instances in which a participant indicates that they have plans to harm themselves or others. This has been specified in the consent document.

In the event a subject expresses suicidal ideation, study staff are trained in a risk of self-harm protocol (uploaded to Zipline). Should a subject endorse the suicidal item on the PHQ-9 assessment or otherwise indicates he/she is actively suicidal during a phone assessment, the Risk of Harm Assessment Procedure (uploaded to Zipline) will be initiated immediately. Should a subject endorse the suicidal item on the PHQ-9 assessment or otherwise indicates he/she is actively suicidal during an online survey, resources will immediately appear on the screen directing the participant to call the Crisis Line, their health care provider, and/or 9-1-1. The study team will be automatically notified and will follow up with the participant according to the Risk of Harm Assessment Procedure. Additionally, staff at the senior living communities have agreed to provide follow up clinical services to any individual identified as at risk of harm. During the consent/assent process, participants are made aware that the study team may share their information with these individuals if there is concern about their safety.

(10.2) Reproductive risks. Are there any risks of the study procedures to men and women (who are subjects, or partner of subjects) related to pregnancy, fertility, lactation or effects on a fetus or neonate?

Examples: direct teratogenic effects; possible germline effects; effects on fertility; effects on a woman's ability to continue a pregnancy; effects on future pregnancies.



→ If no go to question 10.3

→ If yes, answer the following questions:

a. Risks. Describe the magnitude, probability, duration and/or reversibility of the risks.

| | Examples: inform the subjects about the risks and how to minimize them; require a pregnancy test before and during the study; require subjects to use contraception; advise subjects about banking of sperm and ova. |
|---|---|
| | If the use of contraception will be required: describe the allowable methods and the time period when contraception must be used. |
| c. P | Pregnancy. Describe what will be done if a subject (or a subject's partner) becomes pregnant |
| | example; will subjects be required to immediately notify study staff, so that the study procedures can be ontinue or modified, or for a discussion of risks, and/or referrals or counseling? |
| reaction called neph<br>received gadolinium<br>allergic reaction to G<br>a. Describe how the | ent. Answer this question only if the subjects will receive MRI scans. A rare but serious adverse rogenic systemic fibrosis (NSF) has been observed in individuals with kidney disease who based contrast agents (GBCAs) for the scans. Also, a few healthy individuals have a severe iBCAs. The remaining remain |
| · | b. Describe the protocol for handling a severe allergic reaction to the GBCA or any other medical event/emergency during the MRI scan, including who will be responsible for which actions. |
| 10.4 Unforeseeable risks | . Are there any research procedures that may have risks that are currently unforeseeable? |
| Example: using a drug | that hasn't been used before in this subject population. |
| X No | and the outfloating account of the control of the c |
| | es, identify the procedures. |
| patients are under g<br>(supplied for non-res | e under regional or general anesthesiology. Will any research procedures occur while eneral or regional anesthesia, or during the 3 hours preceding general or regional anesthesia search reasons)? |
| | Administration of any drug for research purposes |
| | Inserting an intra-venous (central or peripheral) or intra-arterial line for research purposes |
| | Obtaining samples of blood, urine, bone marrow or cerebrospinal fluid for research purposes |
| Document Date & Version | Researcher Date & Version |

**b. Steps to minimize risk**. Describe the specific steps that will be taken to minimize the

magnitude, probability, or duration of these risks.

| | Obtaining a research sample from tissue or organs that would not otherwise be removed during surgery |
|---|---|
| | Administration of a radio-isotope for research purposes** |
| | Implantation of an experimental device |
| | Other manipulations or procedures performed solely for research purposes (e.g., experimental liver dialysis, experimental brain stimulation) |
| | If any of the boxes are checked: Provide the name and institutional affiliation of a physician anesthesiologist who is a member of the research team or who will serve as a safety consultant about the interactions between the research procedures and the general or regional anesthesia of the subject-patients. If the procedures will be performed at a UW Medicine facility or affiliate, the anesthesiologist must be a UW faculty member, and the Vice Chair of Clinical Research in the UW Department of Anesthesiology and Pain Medicine must be consulted in advance for feasibility, safety and billing. |
| | ** If the box about radio-isotopes is checked: the study team is responsible for informing in advance all appropriate clinical personnel (e.g., nurses, technicians, anesthesiologists, surgeons) about the administration and use of the radio-isotope, to ensure that any personal safety issues (e.g., pregnancy) can be appropriately addressed. This is a condition of IRB approval. |
| by NIH). If required upload the DSMP to | <b>onitoring</b> . A Data and Safety Monitoring Plan (DSMP) is required for clinical trials (as defined for this research, or if there is a DSMP for the research regardless of whether it is required, to <b>Zipline</b> . If it is embedded in another document being uploading (for example, a Study ext box below to name the document that has the DSMP. Alternatively, provide a description text box below. |
| N/A | |
| team members do i | is a double-blinded or single-blinded study in which the participant and/or relevant study not know the group to which the participant is assigned: describe the circumstances under would be necessary, and to whom the un-blinded information would be provided. |
| N/A | |
| withdrawn from the participant, regardl | ticipants. If applicable, describe the anticipated circumstances under which participants will be e research without their consent. Also, describe any procedures for orderly withdrawal of a less of the reason, including whether it will involve partial withdrawal from procedures and ut continued data collection or long-term follow-up. |
| N/A | |

**10.9** Anticipated direct benefits to participants. If there are any direct research-related benefits that some or all individual participants are likely to experience from taking part in the research, describe them below:

Do not include benefits to society or others, and do not include subject payment (if any). Examples: medical benefits such as laboratory tests (if subjects receive the results); psychological resources made available to participants; training or education that is provided.

Test Phase: All older adult participants will receive resources to combat social isolation either through the Stay Connected intervention or the resource sheet provided.

#### (10.10) Return of individual research results.

In this section, provide your plans for the return of individual results. An "individual research result" is any information collected, generated or discovered in the course of a research study that is linked to the identity of a research participant. These may be results from screening procedures, results that are actively sought for purposes of the study, results that are discovered unintentionally, or after analysis of the collected data and/or results has been completed.

See the <u>GUIDANCE Return of Individual Results</u> for information about results that should and should not be returned, validity of results, the Clinical Laboratory Improvement Amendment (CLIA), consent requirements and communicating results.

a. Is it anticipated that the research will produce any individual research results that are clinically actionable?

"Clinically actionable" means that there are established therapeutic or preventive interventions or other available actions that have the potential to change the clinical course of the disease/condition, or lead to an improved health outcome.

In general, every effort should be made to offer results that are clinically actionable, valid and pose life-threatening or severe health consequences if not treated or addressed quickly. Other clinically actionable results should be offered if this can be accomplished without compromising the research.



- $\rightarrow$  If yes, answer the following questions (a.1-a.3).
  - **a.1.** Describe the clinically actionable results that are anticipated and explain which results, if any, could be urgent (i.e. because they pose life-threatening or severe health consequences if not treated or addressed quickly).

Examples of urgent results include very high calcium levels, highly elevated liver function test results, positive results for reportable STDs.

- **a.2.** Explain which of these results will be offered to subjects.
- **a.3.** Explain which results will <u>not</u> be offered to subjects and provide the rationale for not offering these results.

Reasons not to offer the results might include:

- There are serious questions regarding validity or reliability
- Returning the results has the potential to cause bias
- There are insufficient resources to communicate the results effectively and appropriately
- Knowledge of the result could cause psychosocial harm to subjects

| E. | Examples: non-actionable genetic results, clinical tests in the normal range, experimental and/or uncertain results. |
|---|---|
| | X No Yes → If yes, explain which results will be offered to subjects and provide the rationale for |
| | Yes → If yes, explain which results will be offered to subjects and provide the rationale for offering these results. |
| <b>c</b> . D | Describe the validity and reliability of any results that will be offered to subjects. |
| | The IRB will consider evidence of validity such as studies demonstrating diagnostic, prognostic, or predictive value, use of confirmatory testing, and quality management systems. |
| t<br>( | Describe the process for communicating results to subjects and facilitating understanding of the results. In the description, include who will approach the participant with regard to the offer of results, who will communicate the result (if different), the circumstances, timing, and communication methods that will be used. |
| | Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased). |
| t | heck the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form. |
| 5 | See the <b>GUIDANCE Return of Individual Results</b> for information about consent requirements. |
| | Confirmed |
| 10.11 Comm<br>study? | percial products or patents. Is it possible that a commercial product or patent could result from this |
| | No |
| | fes → If yes, describe whether subjects might receive any remuneration/compensation and, if yes, how the amount will be determined. |
| 11 ECONO | OMIC BURDEN TO PARTICIPANTS |
| | al responsibility for research-related injuries. Answer this question only if the lead researcher is <u>not</u> a dent, staff member, or faculty member whose primary paid appointment is at the UW. |
| researcl | n institution involved in conducting the research: Describe who will be financially responsible for h-related injuries experienced by subjects, and any limitations. Describe the process (if any) by which ants may obtain treatment/compensation. |

**b**. Is there a plan for offering subjects any results that are <u>not</u> clinically actionable?

11.2 Costs to subjects. Describe any research-related costs for which subjects and/or their health insurance may be responsible (examples might include: CT scan required for research eligibility screening; co-pays; surgical costs when a subject is randomized to a specific procedure; cost of a device; travel and parking expenses that will not be reimbursed).

N/A

11.3 Reimbursement for costs. Describe any costs to subjects that will be reimbursed (such as travel expenses).

N/A

### **12 RESOURCES**

- 12.1) Faculty Advisor. (For researchers who are students, fellows, or post-docs.) Provide the following information about the faculty advisor.
  - Advisor's name
  - Your relationship with your advisor (for example: graduate advisor; course instructor)
  - Your plans for communication/consultation with your advisor about progress, problems, and changes.
- 12.2 UW Principal Investigator Qualifications. Upload a current or recent Curriculum Vitae (CV), Biosketch (as provided to federal funding agencies), or similar document to the Local Site Documents page in Zipline. The purpose of this is to address the PI's qualifications to conduct the proposed research (education, experience, training, certifications, etc.).

For help with creating a CV, see http://adai.uw.edu/grants/nsf\_biosketch\_template.pdf and https://education.uwmedicine.org/student-affairs/career-advising/year-4/residency-applications/curriculum-vitae/

X The CV will be uploaded.

12.3 UW Study team qualifications. Describe the qualifications and/or training for each <u>UW</u> study team member to fulfill their role on the study and perform study procedures. (You may be asked about non-UW study team members during the review; they should not be described here.) You may list these individuals by name, however if you list an individual by name, you will need to modify this application if that individual is replaced. Alternatively, you can describe study roles and the qualifications and training the PI or study leadership will require for any individual who might fill that role. The IRB will use this information to assess whether risks to subjects are minimized because study activities are being conducted by properly qualified and trained individuals.

Describe: The role (or name of person), the study activities they will perform, and the qualifications or training that are relevant to performing those study activities.

#### **Examples:**

Research Study Coordinator: Obtain consent, administer surveys, blood draw. Will have previous experience coordinating clinical research and be a certified phlebotomist in WA.

<u>Undergraduate Research Assistant:</u> Obtain consent, perform all study procedures. Will have had coursework in research methods, complete an orientation to human subjects protections given by the department, and will receive training from the PI or the graduate student project lead on obtaining consent and debriefing subjects. Acupuncturist: Perform acupuncture procedures and administer surveys. Must be licensed with WA State DoH and complete training in administering research surveys given by the project director, an experienced survey researcher.

<u>Co-Investigator:</u> Supervise MRI and CT scan procedures and data interpretation, obtain consent. MD, specialty in interventional radiology and body imaging. 5-years clinical research experience.

Principal Investigators: Clinical psychologists with extensive experience in the assessment and treatment of depression in diverse populations and in fully remote research

Program Manager: Supervise study team and ensure study procedures are adhered to including consent, assent, and assessment procedures. 3+ year clinical research experience

User Researcher: Complete interviews with older adults & staff members, obtain consent from those groups. 5+ years of user research experience.

Research Study Coordinator: Assist with implementation of all study procedures. Completed CITI trainings in human subjects. 2+ years clinical research experience

Research Study Assistant: Manage scheduling and recruitment inquiries, assist with implementation of all study procedures. Completed CITI training in human subjects research. 1 year clinical research experience.

| 12.4 | <b>12.4 Study team training and communication</b> . Describe how it will be ensured that each study team member is |
|---|---|
| | adequately trained and informed about the research procedures and requirements (including any changes) as |
| | well as their research-related duties and functions. |

There is no study team.

All study team members are required to complete the CITI human subjects and GCP training. Team members are trained on study procedures and changes in formal training sessions, weekly operations and team meetings. New team members are mentored by study PI and staff until they are proficient in their tasks and duties.

# 13 OTHER APPROVALS, PERMISSIONS, and REGULATORY ISSUES

(13.1) Approvals and permissions. Identify any other approvals or permissions that will be obtained. For example: from a school, external site/organization, funding agency, employee union, UW Medicine clinical unit.

Do not attach the approvals and permissions unless requested by the IRB.

We have received permission from participating housing facilities to engage with their staff and residents.

| 13.2 Financial Conflict of Interest. Does any UW member of the team have ownership or other Significant Financial Interest (SFI) with this research as defined by <a href="https://www.uww.nc.nc/months.com/">UW policy GIM 10</a> ? | | |
|---|---|---|
| X No | | |
| Yes | → If yes, has t<br>proposed r | the Office of Research made a determination regarding this SFI as it pertains to the esearch? |
| | No | → If no, contact the Office of Research (206.616.0804, <a href="mailto:research@uw.edu">research@uw.edu</a> ) for guidance on how to obtain the determination |
| | Yes | → If yes, upload the Conflict Management Plan for every UW team member who has a FCOI with respect to the research, to <i>Zipline</i> . If it is not yet available, use the text box to describe whether the Significant Financial Interest has been disclosed |

already to the UW Office of Research and include the FIDS Disclosure ID if available.